# Statistical Analysis Plan: Protocol EBSI-CV-317-004, A Phase 3 Safety, Immunogenicity, and Lot-Consistency Trial of the VLP-Based Chikungunya Vaccine PXVX0317 in Healthy Adults and Adolescents

Version 3.0 20-MAR-2023

ClinicalTrials.gov ID: NCT05072080

# **EMERGENT®**

# Statistical Analysis Plan: Protocol EBSI-CV-317-004, A Phase 3 Safety, Immunogenicity, and Lot-Consistency Trial of the VLP-Based Chikungunya Vaccine PXVX0317 in Healthy Adults and Adolescents

| | | 41 | | | | |
|-----|----|----|---|--------|----|-----|
| Α | 11 | 1 | n | $\cap$ | ۱r | • • |
| / N | u | L | ı | • | " | |

| Statistician | Director,<br>Biostatistics | Signature applied electronically | |
|---|---|---|---|
| Name | Position | Signature | YYYY/MMM/DD |
| Reviewed and Appro | ved: | | |
| Statistical<br>Reviewer | Sr. Director,<br>Biostatistics &<br>Data Sciences | Signature applied electronically | |
| Name | Position | Signature | YYYY/MMM/DD |
| Medical/Scientific<br>Reviewer | Vice President,<br>Clinical<br>Development | Signature applied electronically | |
| Name | Position | Signature | YYYY/MMM/DD |
| Clinical Trial<br>Manager | Sr. Manager,<br>Clinical Trials | Signature applied electronically | |
| Name | Position | Signature | YYYY/MMM/DD |

| <b>Protocol Version</b> | Date |
|-------------------------|-------------|
| Original Protocol 1.0 | 24-AUG-2020 |
| Amendment 2.0 | 06-JUL-2020 |
| Amendment 3.0 | 10-NOV-2021 |
| Amendment 4.0 | 10-FEB-2022 |
| Amendment 5.0 | 20-MAR-2023 |
| SAP Version | Date |
| 1.0 (Final) | 27-OCT-2020 |
| 2.0 (Final) | 22-JUL-2021 |
| 3.0 (Final) | 20-MAR-2023 |

## **Summary of Changes**

| Version | Summary of Major Change(s) and Impact | <b>Revision Date</b> |
|---|---|---|
| Version<br>1.0 | First approved version of SAP. | 27-OCT-2020 |
| Version 2.0 | Updated to correspond to Protocol Amendment 2.0 (addition of Day 15, removal of success criterion at Day 8, and change to hierarchical secondary endpoint strategy). | 22-JUL-2021 |
| Version 3.0 | Made minor edits for consistency. Added MAAEs throughout. Removed statement that randomization number is hidden. Updated coding dictionary versions. Added clarification that participants missing Day 1 SNA are excluded from IEP. Updated for alignment with protocol version 5.0: changed threshold to added backup paper memory aid (diary), removed references to FDA and EMA, removed hierarchy on coprimary endpoints, designated hierarchical secondary endpoints as key, added success criterion at Day 15, simplified the "other titers" secondary endpoint to ≥15 and 4-fold rise only, added EMA definition of seroresponse rate as the presumptive seroprotection rate, and updated "CHIKV-luc assay anti-CHIKV SNA NT <sub>80</sub> " to "anti-CHIKV human SNA assay." Added analysis visit windows for SNA to mitigate the risk of data entered in an incorrect visit in the database. Updated Appendix I TFL list to align with that for study -005. Added specification for listing of participants not meeting randomization criteria to be programmed from protocol deviations and not (original) entry criteria CRF. Added new AESI table including solicited events, added age strata to selected AE tables, and added new listing of AEs during acute observation period. Removed Appendix III and text referring to MedDRA SMQ. Excluded from tables solicited events starting after Day 8 and those AEs starting past Day 29 that are not SAEs, AESI, or MAAEs. Excluded postdose vital signs fever from solicited AEs. Added discussion of screen failure participants and empty participant identifiers. | 20-MAR-2023 |

#### **Table of Contents**

| 1 | INT | RODUCTION | 9 |
|---|---|---|---|
| 2 | PRC | OTOCOL SUMMARY | 9 |
| | 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.2<br>2.3<br>2.3.1<br>2.3.2<br>2.3.3 | Exploratory Objectives Study Design and Conduct Randomization and Blinding Method of Randomization | 9<br>10<br>15<br>15 |
| 3 | STU | DY ENDPOINTS | 16 |
| | 3.1.1<br>3.1.2<br>3.1.3<br>3.2<br>3.3<br>3.4<br>3.5 | $\mathcal{L}$ | 1617171717 |
| 4 | POV | VER AND SAMPLE SIZE CONSIDERATIONS | 18 |
| | 4.1<br>4.2<br>4.3 | Sample Size and Power for Immunogenicity | 18 |
| 5 | DAT | TA CONSIDERATIONS | 19 |
| | 5.1.1 5.1.2 5.2.1 5.2.2 5.3 | Protocol Deviations Important Deviations Reporting of Protocol Deviations Analysis Populations | 1919192020 |
| | 5.4<br>5.5 | Analysis Groups | 21 |
| | 5.6<br>5.7<br>5.8 | Definition of Baseline | 22 |
| 6 | 5.9 | Adverse Event Toxicity/Severity Grading TISTICAL CONSIDERATIONS | 22 |

| | 6.1 | Statistical Considerations | 23 |
|---|---|---|---|
| | 6.1.1 | Seroresponse Rates | 23 |
| | 6.1.2 | Geometric Mean Titers and Geometric Mean Fold Increase | 24 |
| | <b>6.2</b> | Units and Precision | 24 |
| | 6.3 | Derived Variables | 25 |
| | <b>6.4</b> | Statistical Hypotheses | |
| | 6.4.1 | Coprimary Immunogenicity Endpoints | 28 |
| | 6.4.2 | Key Secondary Immunogenicity Endpoints | |
| | 6.5 | Handling of Missing Data and Other Data Issues | 30 |
| | 6.5.1 | Missing or Partial Dates for Solicited Adverse Events | 30 |
| | 6.5.2 | Missing or Partial Dates for Unsolicited Adverse Events and Concomitant | |
| | | Medications | |
| | 6.5.3 | Missing Outcome and Covariates | |
| | 6.5.4 | Non-Quantifiable Laboratory Data | |
| | 6.5.5 | Implausible Participant Reported Outcomes | |
| | 6.6 | Adjustment for Covariates | |
| | <b>6.7</b> | Multicenter Study | |
| | <b>6.8</b> | Subgroup Analysis | |
| | 6.9 | Multiplicity Adjustment | |
| | 6.9.1 | Coprimary Immunogenicity Endpoints | 32 |
| | 6.9.2 | Key Secondary Immunogenicity Endpoints | 32 |
| 7 | STU | DY POPULATION CHARACTERISTICS | 33 |
| | | | 22 |
| | <b>7.1</b> | Participant Disposition | <b>ა</b> : |
| | 7.1<br>7.2 | Participant Disposition Protocol Deviations | |
| 8 | 7.2 | | 33 |
| 8 | 7.2<br>IMN | Protocol Deviations IUNOGENICITY ANALYSIS | 33 |
| 8 | 7.2<br>IMM<br>8.1 | Protocol Deviations IUNOGENICITY ANALYSIS Populations Analyzed | 33<br>33 |
| 8 | 7.2<br>IMM<br>8.1<br>8.2 | Protocol Deviations | 33<br>33 |
| 8 | 7.2<br>IMM<br>8.1<br>8.2<br>8.2.1 | Protocol Deviations IUNOGENICITY ANALYSIS Populations Analyzed Demographics and Baseline Characteristics Demographics | 33<br>33<br>34 |
| 8 | 7.2<br>IMM<br>8.1<br>8.2<br>8.2.1<br>8.2.2 | Protocol Deviations IUNOGENICITY ANALYSIS Populations Analyzed Demographics and Baseline Characteristics Demographics Baseline Disease Characteristics. | 33<br>33<br>34<br>34 |
| 8 | 7.2<br>IMM<br>8.1<br>8.2<br>8.2.1 | Protocol Deviations IUNOGENICITY ANALYSIS Populations Analyzed Demographics and Baseline Characteristics Demographics Baseline Disease Characteristics Medical History | 33<br>34<br>34<br>34 |
| 8 | 7.2<br>IMM<br>8.1<br>8.2<br>8.2.1<br>8.2.2<br>8.2.3 | Protocol Deviations IUNOGENICITY ANALYSIS Populations Analyzed Demographics and Baseline Characteristics Demographics Baseline Disease Characteristics Medical History Prior and Concomitant Medications and Vaccines | 33<br>33<br>34<br>34<br>34 |
| 8 | 7.2<br>IMM<br>8.1<br>8.2<br>8.2.1<br>8.2.2<br>8.2.3<br>8.2.4 | Protocol Deviations IUNOGENICITY ANALYSIS Populations Analyzed Demographics and Baseline Characteristics Demographics Baseline Disease Characteristics Medical History Prior and Concomitant Medications and Vaccines Treatment Compliance | 33<br>34<br>34<br>34<br>34<br>34 |
| 8 | 7.2<br>IMM<br>8.1<br>8.2<br>8.2.1<br>8.2.2<br>8.2.3<br>8.2.4<br>8.3 | Protocol Deviations IUNOGENICITY ANALYSIS Populations Analyzed Demographics and Baseline Characteristics Demographics Baseline Disease Characteristics Medical History Prior and Concomitant Medications and Vaccines Treatment Compliance Immunogenicity Analysis | 33<br>34<br>34<br>34<br>34<br>34 |
| 8 | 7.2<br>IMM<br>8.1<br>8.2<br>8.2.1<br>8.2.2<br>8.2.3<br>8.2.4<br>8.3<br>8.4 | Protocol Deviations IUNOGENICITY ANALYSIS Populations Analyzed Demographics and Baseline Characteristics Demographics Baseline Disease Characteristics Medical History Prior and Concomitant Medications and Vaccines Treatment Compliance | 33<br>33<br>34<br>34<br>34<br>34<br>34<br>35 |
| 8 | 7.2<br>IMM<br>8.1<br>8.2<br>8.2.1<br>8.2.2<br>8.2.3<br>8.2.4<br>8.3<br>8.4<br>8.4.1 | Protocol Deviations IUNOGENICITY ANALYSIS Populations Analyzed Demographics and Baseline Characteristics Demographics Baseline Disease Characteristics Medical History Prior and Concomitant Medications and Vaccines Treatment Compliance Immunogenicity Analysis Coprimary Immunogenicity Endpoints | 33<br>33<br>34<br>34<br>34<br>35<br>35 |
| 8 | 7.2 IMN 8.1 8.2 8.2.1 8.2.2 8.2.3 8.2.4 8.3 8.4 8.4.1 8.4.2 | Protocol Deviations IUNOGENICITY ANALYSIS Populations Analyzed Demographics and Baseline Characteristics Demographics Baseline Disease Characteristics Medical History Prior and Concomitant Medications and Vaccines Treatment Compliance Immunogenicity Analysis Coprimary Immunogenicity Endpoints Secondary Immunogenicity Endpoints | 33<br>33<br>34<br>34<br>34<br>35<br>36<br>36 |
| 9 | 7.2 IMN 8.1 8.2 8.2.1 8.2.2 8.2.3 8.2.4 8.3 8.4 8.4.1 8.4.2 8.4.3 8.5 | Protocol Deviations IUNOGENICITY ANALYSIS Populations Analyzed Demographics and Baseline Characteristics Demographics Baseline Disease Characteristics Medical History Prior and Concomitant Medications and Vaccines Treatment Compliance Immunogenicity Analysis Coprimary Immunogenicity Endpoints Secondary Immunogenicity Endpoints Exploratory Immunogenicity Endpoints | 33<br>33<br>34<br>34<br>34<br>35<br>36<br>38<br>38 |
| | 7.2 IMN 8.1 8.2 8.2.1 8.2.2 8.2.3 8.2.4 8.3 8.4 8.4.1 8.4.2 8.4.3 8.5 | Protocol Deviations IUNOGENICITY ANALYSIS Populations Analyzed Demographics and Baseline Characteristics Demographics Baseline Disease Characteristics Medical History Prior and Concomitant Medications and Vaccines Treatment Compliance Immunogenicity Analysis Coprimary Immunogenicity Endpoints Secondary Immunogenicity Endpoints Exploratory Immunogenicity Endpoints Exploratory Immunogenicity Endpoints Pharmacokinetic and Pharmacodynamic Analysis | 33<br>33<br>34<br>34<br>34<br>35<br>36<br>38<br>38 |
| | 7.2 IMM 8.1 8.2 8.2.1 8.2.2 8.2.3 8.2.4 8.3 8.4 8.4.1 8.4.2 8.4.3 8.5 SAF | Protocol Deviations IUNOGENICITY ANALYSIS | 3333343434353538383838 |
| | 7.2 IMM 8.1 8.2 8.2.1 8.2.2 8.2.3 8.2.4 8.3 8.4 8.4.1 8.4.2 8.4.3 8.5 SAF | Protocol Deviations IUNOGENICITY ANALYSIS Populations Analyzed Demographics and Baseline Characteristics Demographics Baseline Disease Characteristics Medical History Prior and Concomitant Medications and Vaccines Treatment Compliance Immunogenicity Analysis Coprimary Immunogenicity Endpoints Secondary Immunogenicity Endpoints Exploratory Immunogenicity Endpoints Pharmacokinetic and Pharmacodynamic Analysis Extent of Exposure Adverse Events Overall Summary of Solicited and Unsolicited Adverse Events | 333434343435353838383838 |
| | 7.2 IMM 8.1 8.2 8.2.1 8.2.2 8.2.3 8.2.4 8.3 8.4 8.4.1 8.4.2 8.4.3 8.5 SAF | Protocol Deviations IUNOGENICITY ANALYSIS | 33333434343435353638383838 |

| 9.3 | Deaths, Other Serious Adverse Events and Other Significant Adverse | |
|---|---|---|
| 9.3.1 | | |
| 9.3.2 | | 40 |
| 9.3.3 | Adverse Event of Special Interest from Day 1 to Day 183 End of Study | |
| | Visit | 40 |
| 9.3.4 | | |
| | | 41 |
| 9.3.5 | | |
| 9.5.2 | Physical Examinations | 41 |
| DAT | TA MONITORING AND INTERIM ANALYSIS | 42 |
| 10.1 | Safety Monitoring Committee | 42 |
| 10.2 | | |
| REE | TERENCES | 43 |
| ILLI | | 10 |
| | Appendices | |
| PEND | IX I LIST OF TABLES, FIGURES AND LISTINGS | 44 |
| PEND | IX II TOXICITY GRADING SCALE | 48 |
| | 9.3.1<br>9.3.2<br>9.3.3<br>9.3.4<br>9.3.5<br>9.3.6<br><b>9.4</b><br>9.4.2<br><b>9.5</b><br>9.5.1<br>9.5.2<br><b>DAT</b><br><b>10.1</b><br><b>10.2</b><br><b>REF</b> | Events 9.3.1 Deaths from Day 1 to Day 183 End of Study Visit 9.3.2 Serious Adverse Events from Day 1 to Day 183 End of Study Visit 9.3.3 Adverse Event of Special Interest from Day 1 to Day 183 End of Study Visit 9.3.4 Medically Attended Adverse Events from Day 1 to Day 183 End of Study Visit 9.3.5 Adverse Events Leading to Study Discontinuation from Day 1 to Day 183 End of Study Visit 9.3.6 Day 1 Adverse Events 9.4 Clinical Laboratory Tests 9.4.1 Pregnancy Testing 9.4.2 Viral Serology Testing at Screening 9.5 Vital Signs, Physical Findings and Other Variables Related to Safety 9.5.1 Vital Signs 9.5.2 Physical Examinations DATA MONITORING AND INTERIM ANALYSIS 10.1 Safety Monitoring Committee 10.2 Interim Analysis REFERENCES. |

#### PXVX0317 Vaccine EBSI-CV-317-004 SAP

## **List of Figures**

| Figure 1 | EBSI-CV-317-004 Schematic Diagram of Study Design | 12 |
|----------|---------------------------------------------------|----|
| _ | Schedule of Events. | |

#### List of Abbreviations and Definition of Terms

AE Adverse Event

AESI Adverse Events of Special Interest

ANCOVA Analysis of Covariance
ANOVA Analysis of Variance

ATC Anatomic Therapeutic Chemical classification

BMI Body Mass Index
CI Confidence Interval
CHIKV Chikungunya Virus
CSR Clinical Study Report

eCRF Electronic Case Report Form

e-diary Electronic Diary

EDC Electronic Data Capture
EMA European Medicines Agency

EOS End of Study Visit

FDA Food and Drug Administration
FSH Follicle-Stimulating Hormone
GMFI Geometric Mean Fold Increase

GMT Geometric Mean Titer
HBsAg Hepatitis B surface antigen

HBV Hepatitis B Virus HCV Hepatitis C Virus

HIV Human Immunodeficiency Virus

ICF Informed Consent Form

ICH International Conference on Harmonisation
IEP Immunogenicity Evaluable Population

IM Intramuscular

IP Investigational Product

LLOQ Lower Limit of Quantification

MAAE Medically attended adverse event

MedDRA Medical Dictionary for Regulatory Activities

mITT Modified Intent-to-Treat

mL milliliter(s) mm millimeter(s)

NT<sub>80</sub> 80% Neutralizing Titer

PT Preferred Term

PXVX0317 Vaccine Investigational Product

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SD Standard Deviation

# PXVX0317 Vaccine EBSI-CV-317-004 SAP

SDTM Standard Data Tabulation Model
SMC Safety Monitoring Committee
SNA Serum Neutralizing Antibody

SOC System Organ Class

TFL Tables, Figures, and Listings

US United States
VLP Virus-like Particle

WHO World Health Organization

#### 1 INTRODUCTION

This Statistical Analysis Plan (SAP) is based on Protocol EBSI-CV-317-004, "A Phase 3 Safety, Immunogenicity, and Lot-Consistency Trial of the VLP-Based Chikungunya Vaccine PXVX0317 in Healthy Adults and Adolescents" (Version 5.0 date 20-MAR-2023). This document specifies details of the definitions of the derived variables, analysis methods, assumptions and data handling conventions. The document is accompanied by mock-up tables, figures, and listings (TFL shells). Some further details on the calculation of derived variables are provided as programmer's notes in the TFL shells. The TFL shells serve only as a guide for programming the final TFL. They are working documents and can be updated as needed.

#### 2 PROTOCOL SUMMARY

#### 2.1 Study Objectives

#### 2.1.1 Coprimary Objectives

- To evaluate the safety of PXVX0317 in healthy adult and adolescent participants 12 to <65 years of age.
- To compare the anti-chikungunya virus (CHIKV) serum neutralizing antibody (SNA) response to PXVX0317 and placebo at Day 22, as measured by geometric mean titer (GMT) and clinically relevant difference in seroresponse rate (PXVX0317 minus placebo).

**Note:** Seroresponse rate (considered the presumptive seroprotection rate) is defined as the percentage of participants who achieve an anti-CHIKV SNA titer

• To demonstrate the consistency of the anti-CHIKV SNA response across three consecutively manufactured lots of PXVX0317 at Day 22 as measured by GMT.

#### 2.1.2 Secondary Objectives

- To compare the anti-CHIKV SNA response to PXVX0317 and placebo at Day 15, Day 183, and Day 8, as measured by GMT and seroresponse rate.
- To compare the anti-CHIKV SNA response to PXVX0317 and placebo in participants 12 to <18 years of age, participants 18 to <46, and participants 46 to <65 years of age as measured by GMT and seroresponse rate.

#### 2.1.3 Exploratory Objectives

 To evaluate anti-CHIKV SNA response across three consecutively manufactured lots of PXVX0317 as measured by seroresponse rate for each lot at Day 22 in participants 18 to <46 years of age.</li>

#### 2.2 Study Design and Conduct

This is a phase 3 randomized, placebo-controlled, double-blind, parallel-group design with four treatment groups. Participants are randomized in a 2:2:2:1 ratio within each of the three age strata (ages 12 to <18, 18 to <46, and 46 to <65) to receive one of three consecutively manufactured lots of PXVX0317 or placebo. With 3150 participants enrolled, the treatment group totals are estimated as follows:

- Group 1- PXVX0317 lot A: n=900
- Group 2- PXVX0317 lot B: n=900
- Group 3- PXVX0317 lot C: n=900
- Group 4- Placebo: n=450

A nested lot consistency sub study is performed in adult participants 18 to <46 years of age in the PXVX0317 treatment groups (lot A, lot B, and lot C).

This multicenter study is conducted in the US, using approximately 50 sites. At least 3150 healthy US adolescent and adult participants ages 12 to <65 are enrolled, stratified in three age groups: 12 to <18, 18 to <46, and 46 to <65 years of age. Enrollment targets at least 245 participants (210 PXVX0317 and 35 placebo participants) into the youngest and oldest age groups (12 to <18 and 46 to <65 years of age, respectively). The middle age group must include at least 1050 participants to provide adequate power for the lot consistency analysis.

The per participant estimated total study duration is 212 days. The screening window is no greater than 30 days prior to Day 1 (randomization and administration of investigational product [IP]). Screening assessments include informed consent (and assent for adolescent participants 12 to <18 years of age), review of eligibility criteria, medical history, prior and concomitant medications, demography, physical examination including height and weight for body mass index calculation, vital signs, follicle-stimulating hormone (FSH) or serum pregnancy test for female participants, urine toxicology screening per investigator's discretion and viral markers for hepatitis B surface antigen (HBsAg), hepatitis C (HCV) and human immune deficiency virus 1 and 2 (HIV-1/HIV-2).

Prior to IP administration on Day 1 (baseline), eligibility, medical history and concomitant medications are reviewed, and a baseline anti-CHIKV SNA sample are drawn. Urine pregnancy test is performed at Day 1 before IP administration for women of childbearing potential. Vital signs including blood pressure, heart rate, respiratory rate and temperature are taken on Day 1 before and after IP administration. Directed physical examinations are performed if indicated at Days 1, 8, 15, 22 and Day 183 End of Study Visit (EOS). The immune response to PXVX0317 is measured by anti-CHIKV SNA at Day 8, Day 15, Day 22 (coprimary endpoints are at Day 22) and Day 183 EOS (or at Early Discontinuation/Withdrawal). No safety laboratory samples are collected as part of the study.

Solicited adverse events (AEs) are collected from IP administration until Day 8 using an electronic diary (e-diary) or backup paper diary. Severity and relationship of solicited AEs are assessed by the investigator in the same manner as unsolicited AEs. Unsolicited AEs (AEs not listed in the diary) are collected from Day 1 through 28 days post-vaccination. Serious adverse events (SAEs), adverse events of special interest (AESI; see Section 6.3 for

definition), and medically attended AEs (MAAEs) are collected for all participants from Day 1 through Day 183 EOS. Telephonic visits occur at Days 29 and 92 to evaluate unsolicited AEs (Day 29 only), MAAEs, SAEs, and AESI and to review concomitant medications.

An independent Safety Monitoring Committee (SMC) reviews aggregated, blinded safety data after the 300<sup>th</sup> enrolled participant passes Day 29, and again after the last enrolled participant passes Day 29.

Refer to Figure 1, Schematic Diagram of Study Design, and Figure 2, Schedule of Events.



Figure 1 EBSI-CV-317-004 Schematic Diagram of Study Design

Figure 2 **Schedule of Events** 

| | Screening<br>Visit 1 | Day 1<br>Visit 2 | Day 8<br>Visit 3 | Day 15<br>Visit 4 | Day 22<br>Visit 5 | Day 29<br>Visit 6<br>(Phone) | Day 92<br>Visit 7<br>(Phone) | Day 183 <sup>13</sup><br>Visit 8 |
|---|---|---|---|---|---|---|---|---|
| Window (days) | Within 30 days<br>of Day 1 | | -1/+3 | -1/+3 | -1/+3 | ±1 | ±3 | -14/+7 |
| Informed Consent/Assent | X | | | | | | | |
| Eligibility Criteria | X | *X | | | | | | |
| Medical History | $X^1$ | *X <sup>2</sup> | | | | | | |
| Demography | X | | | | | | | |
| Physical Exam | $X^3$ | *X <sup>4</sup> | X <sup>4</sup> | X <sup>4</sup> | X <sup>4</sup> | | | X <sup>4</sup> |
| Viral Marker testing (HIV-1/2, anti-HCV <sup>5</sup> , HBsAg) | X | | | | | | | |
| Urine Toxicology <sup>6</sup> | X | | | | | | | |
| Vital Signs <sup>7</sup> | X | *X <sup>8</sup> | | | | | | |
| Pregnancy Test (female of CBP) | X <sup>9</sup> | *X <sup>10</sup> | | | | | | |
| FSH Levels (post-menopausal female) | X | | | | | | | |
| Randomization | | *X | | | | | | |
| Administration of Investigational Product | | X | | | | | | |
| Acute Observation | | X | | | | | | |
| Solicited AEs | | X | X | | | | | |
| Unsolicited AEs | | X | X | X | X | X | | |
| SAEs | | X | X | X | X | X | X | X |
| AESI | | X | X | X | X | X | X | X |
| MAAE | | X | X | X | X | X | X | X |
| Concomitant Medications | X | X | X | X | X | X | $X^{11}$ | $X^{11}$ |
| Anti-CHIKV SNA Sample | | *X | X | X | X | | | X |
| e-Diary Training and Distribution of Devices <sup>12</sup> | | X | | | | | | |
| e-Diary Collection and Review | | | X | | | | | |

<sup>\*</sup>To be done prior to IP administration. FSH = follicle stimulating hormone

<sup>&</sup>lt;sup>1</sup>To include presence of joint pain.

<sup>&</sup>lt;sup>2</sup>To be updated if necessary.

<sup>&</sup>lt;sup>3</sup>Complete physical exam.

<sup>&</sup>lt;sup>4</sup>Directed physical exam, as needed.

<sup>&</sup>lt;sup>5</sup>If HCV antibody is positive HCV ribonucleic acid (RNA) testing can be performed.

<sup>&</sup>lt;sup>6</sup>Urine toxicology, per investigator's discretion.

<sup>&</sup>lt;sup>7</sup>To include height and body weight (for BMI calculation).

<sup>&</sup>lt;sup>8</sup>To be taken before and after IP administration.

<sup>&</sup>lt;sup>9</sup>Serum pregnancy test.

<sup>&</sup>lt;sup>10</sup>Urine pregnancy test.

<sup>&</sup>lt;sup>11</sup>Concomitant medications associated with SAE/AESI/MAAE only.

<sup>&</sup>lt;sup>12</sup>Smart phone (e-diary), digital thermometer, and ruler.

<sup>&</sup>lt;sup>13</sup>Early Discontinuation/Withdrawal Visit occurring within 7 days postvaccination, from 7 to 21 days postvaccination, or ≥22 days postvaccination the Visit 3, Visit 5, or Visit 8 schedule will be followed respectively.

#### 2.3 Randomization and Blinding

#### 2.3.1 Method of Randomization

Participants are randomized on Day 1 following confirmation of eligibility and immediately prior to IP administration. Study personnel randomize the participant within the electronic data capture (EDC) system, and a randomization number is generated from the EDC randomization module. The EDC randomization module matches the randomization number to an IP kit available at the site and inform the study personnel of the assigned kit. Study personnel use the appropriate kit for administration to the participant.

Participants are considered enrolled once a randomization number has been assigned within the EDC system. The study is conducted as a double-blind study through Day 183 EOS. The participants, site personnel (including the investigator) and the Sponsor do not know participants' individual treatment assignments until all participants have completed their participation in the study through the Day 183 EOS and the database has been cleaned and locked

#### 2.3.2 Randomization Errors

A *misrandomization* is defined as a participant receiving a study treatment other than the one assigned by randomization.

A *stratification error* occurs when a participant is randomized based on incorrect stratification information at Day 1 (baseline) or if a participant is mistakenly put into a wrong block.

In either case, the participant uses up one position in the assigned block and randomization continues. Both misrandomization and stratification errors are reported as protocol deviations.

#### 2.3.3 Blinding and Unblinding

Study participants, the investigator, and study site personnel remain blinded to all randomization assignments throughout the study. Sponsor's Medical Monitor and personnel who are in regular contact with the study site and/or involved with documentation associated with the study remain blinded to all participant randomization assignments.

The following safeguards are employed to reduce the risk of inadvertent unblinding:

- Use of a standardized pre-filled syringe and injection volume for all injections.
- All PXVX0317 and placebo syringes have a semi-transparent barrel cover to mask any difference in appearance between placebo and PXVX0317.
- No Sponsor personnel has access to the randomization schedule. No site personnel has
  access to treatment assignments. The Randomization and Trial Supply Management
  component of the vendor EDC system allows for unblinding of individual participants in
  an emergency by the investigator. The investigator must attempt to notify the Sponsor's
  Medical Monitor prior to unblinding and must notify the Medical Monitor within

24 hours after unblinding at the latest. If the investigator is unable to access the vendor EDC system, then the Medical Monitor may assist by calling the vendor EDC helpline for emergency unblinding. Emergency unblinding is documented as a protocol deviation.

- Assays are run in a blinded manner. The assay titer results are not delivered to the Sponsor data management and analysis team until after database lock, as they are potentially unblinding.
- Should any participant or site personnel become inadvertently unblinded, the investigator promptly (within 24 hours of their awareness of the error) discloses the event to the Sponsor's Medical Monitor in a blinded fashion (disclosing only participant number, not treatment) so that corrective action can be initiated. The unblinding sequence of events is documented and retained as source documents. A protocol deviation is entered in the electronic case report form (eCRF).

Refer to the separate Blind Maintenance Plan for further details.

An individual participant is considered to have completed study participation after completion of the Day 183 EOS and any required safety follow-up. Upon completion of the study for all participants, the study database is cleaned and locked per the Sponsor's standard operating procedures. Unblinding occurs per the Sponsor's standard operating procedures after the SAP is finalized and approved and the database is locked. The Sponsor completes an unblinding request form, approved by the study statistician and medical/scientific reviewer and sends the completed and approved form to the EDC vendor to request release of the randomization assignments to the Sponsor for final analysis.

#### 3 STUDY ENDPOINTS

#### 3.1 Immunogenicity Endpoints

#### 3.1.1 Coprimary Immunogenicity Endpoints

• Difference in anti-CHIKV SNA seroresponse rate (PXVX0317 minus placebo) and associated 95% confidence interval (CI) at Day 22.

**Note:** Seroresponse rate (considered the presumptive seroprotection rate) is defined as the percentage of participants who achieve an anti-CHIKV SNA titer

• Anti-CHIKV SNA GMT and associated 95% CIs at Day 22 for PXVX0317 and placebo.

Each endpoint is summarized for all age strata pooled and for individual age strata, as well as by sex and by race group (white and non-white) and ethnicity group (Hispanic or Latino and Not Hispanic or Latino).

• Anti-CHIKV SNA GMT ratio with associated 95% CIs between all three pairs of PXVX0317 lots (A:B, A:C, B:C) (adults 18 to <46 years of age) at Day 22.

Note that success on the Day 22 lot consistency endpoint is only required for FDA.

#### 3.1.2 Secondary Immunogenicity Endpoints

- **Key Secondary Endpoints:** Difference in anti-CHIKV SNA seroresponse rate (PXVX0317 minus placebo) with associated 95% CI at Day 15, Day 183, and Day 8, in that order.
- Anti-CHIKV SNA GMTs by study arm with associated 95% CIs at Day 8, Day 15, and Day 183.
- Geometric mean fold increase (GMFI) in anti-CHIKV SNA titer from baseline (Day 1) to Days 8, 15, 22 and 183.
- Number and percentage of participants with an anti-CHIKV SNA titer ≥15 and 4-fold rise over baseline at Days 8, 15, 22 and 183.

Each endpoint is summarized for all age strata pooled and for individual age strata.

- If the baseline seropositive (anti-CHIKV SNA titer ≥LLOQ) rate is ≥10%: Difference in anti-CHIKV SNA composite seroresponse rate (PXVX0317 minus placebo) and associated 95% CI at Day 22. The composite seroresponse rate endpoint is defined as follows:
  - For participants seronegative at baseline (anti-CHIKV SNA titer <LLOQ), a seroresponse is defined as an anti-CHIKV SNA titer at Day 22.
  - For participants seropositive at baseline (anti-CHIKV SNA titer ≥LLOQ), a seroresponse is defined as ≥4-fold rise from Day 1 (baseline) in anti-CHIKV SNA titer at Day 22.
- If the baseline seropositive (anti-CHIKV SNA titer ≥LLOQ) rate is ≥10%: Difference between anti-CHIKV SNA GMT and associated 95% CIs at Day 22 for PXVX0317 and placebo, where baseline log-transformed SNA assay titer is a covariate in the analysis of covariance (ANCOVA) model.

Each endpoint is summarized for all age strata pooled and for individual age strata.

#### 3.1.3 Exploratory Immunogenicity Endpoints

 Anti-CHIKV SNA seroresponse rate difference with associated 95% CIs for each pair of PXVX0317 lots (A minus B, A minus C, B minus C) (adults 18 to <46 years of age) at Day 22.

#### 3.2 Safety Endpoints

- Incidence of solicited AEs through Day 8 for PXVX0317 and placebo.
- Incidence of unsolicited AEs through Day 29 for PXVX0317 and placebo.
- Incidence of AESI and SAEs and MAAEs through Day 183 for PXVX0317 and placebo.

#### 3.3 Pharmacokinetic Endpoints

Not applicable.

#### 3.4 Pharmacodynamics Endpoints

Not applicable.

#### 3.5 Exploratory Endpoints

See Section 3.1.3.

#### 4 POWER AND SAMPLE SIZE CONSIDERATIONS

#### 4.1 Sample Size and Power for Immunogenicity

The statistical comparison between the PXVX0317 and placebo treatment groups is based on the difference between treatment groups in seroresponse rate (percentage of participants with anti-CHIKV titer as measured by the human SNA assay) at Day 22, which is tested using a chi-square test with a two-sided alpha=0.05 in the immunogenicity evaluable population (IEP) across all age groups combined. The analysis is repeated for the modified intent-to-treat population (mITT) as a measure of the robustness of the result.

Based on the data from the phase 2 study (protocol PXVX-CV-317-001), the seroresponse rate for PXVX0317 vaccine is expected to be approximately vs <5% for the placebo participants at Day 22. With an assumed 10% rate of non-evaluable participants, the power to show superiority over placebo with 2430 PXVX0317 vaccine and 405 placebo evaluable participants is >99.9% for the combined ages groups. The power is 99% for each of the smaller 12 to <18 and 46 to <65 age groups with samples sizes of 189 vs 32 evaluable participants (PXVX0317: placebo).

The difference in seroresponse rate between PXVX0317 and placebo groups that is considered clinically relevant is With 2430 PXVX0317-treated participants and a target seroresponse rate of vs a rate of 0% for placebo, the width of a two-sided 95% CI would be  $\pm 1.2\%$ . The difference in seroresponse rate must be above for the lower bound of the 95% CI for the difference to be

#### 4.2 Sample Size and Power for Lot Consistency

The second consideration for sizing the study is ensuring adequate power for the lot consistency equivalence intervals testing immunogenicity at Day 22, as measured by anti-CHIKV SNA GMT ratios between all three pairs of consecutively manufactured PXVX0317 lots (A:B, A:C, B:C) in the 18 to <46 years of age stratum for the IEP. Pairwise testing of lots is performed without multiplicity adjustment, and for each GMT ratio the two-sided 95% CI must fall within the equivalence interval of [0.667, 1.5] for the lots to be considered equivalent.

On the log<sub>10</sub> scale, two one-sided equivalence tests have 95% power to reject the null hypothesis that the difference in mean titers between lots is below -0.176 or above 0.176 in favor of an alternative hypothesis of equivalence when the expected difference in log<sub>10</sub> means is 0, the common standard deviation (SD) is 0.455, each test is at the 2.5% level and the sample size in each lot is 207. The SD estimate was based on the upper bound of an

80% CI on the SD on the log<sub>10</sub> scale observed in the anti-CHIKV human SNA assay on samples collected 4 weeks after participants were treated with a single dose of PXVX0317. To be conservative, at least 1050 evaluable participants (300 participants in each lot along with 150 placebo participants) need to be enrolled into the 18 to <46 age group to provide adequate power for the lot consistency objective.

#### 4.3 Sample Size and Power for Adverse Events

The final consideration for the sample size of the study is the size of the pre-licensure safety database. With 2700 participants receiving any lot of PXVX0317, this study is 93.3% likely to detect at least one AE with a true frequency of  $\geq 0.1\%$  (i.e., "uncommon").

#### 5 DATA CONSIDERATIONS

#### 5.1 Participant Screening

#### 5.1.1 Screen Failure Participants

A note to file was generated for this study to document that no data collection conventions were prespecified for screen failure participants. The only data domains considered necessary for screen failure participants are demographics, eligibility criteria, and disposition data.

#### 5.1.2 Rescreening and Empty Participant Identifiers

The study protocol states that rescreened participants should use the original participant identifier. However, in some cases, sites rescreened participants with a new participant identifier number. Once data were consolidated for rescreened participants into the participant identifier used for randomization, an empty participant identifier resulted. In other cases, extra participant identifier numbers were generated inadvertently. These blank identifiers were not deleted from the study database for technical reasons. A note to file was written for this study to specify that participant identifiers empty of data (i.e., blank participant IDs) would not be mapped to SDTM nor included in any clinical study report analyses.

#### **5.2** Protocol Deviations

A deviation occurs when site personnel or a participant does not adhere to the protocol's stipulated requirements, whether inadvertently or planned. All identified protocol deviations are documented (entered by the monitor in EDC) and classified by category and type (important/not important). In addition, nonoverlapping programmatic checks for protocol deviations are run by both the Sponsor and the EDC vendor. Programmatically identified protocol deviations are also entered/uploaded to the EDC and classified by category and type (important/not important).

#### 5.2.1 Important Deviations

Important protocol deviations are defined by ICH E3 (ICH, 1996) as those "that might significantly affect the completeness, accuracy, and/or reliability of the study data or that might significantly affect a participant's rights, safety, or well-being". Examples of important protocol deviations include:

- Participants who were enrolled/randomized but did not meet study eligibility criteria.
- Participants randomized but not treated.
- Participants with misrandomization or stratification errors.
- Participants who received a prohibited prior or concomitant medication or vaccine.
- Participants who previously received an investigational CHIKV vaccine/product, including but not limited to prior vaccination in EBSI-CV-317-004.
- Other deviations from key study procedures such as accidental unblinding or participant noncompliance with assessment of primary outcome measures (e.g., missing serum samples, significantly out of window assessments).

#### **5.2.2** Reporting of Protocol Deviations

All protocol deviations are contained in the Study Data Tabulation Model (SDTM) datasets. Protocol deviations assessed as important are tabulated by treatment group and listed by participant for the randomized population (see Section 7.2).

Deviations excluding participants from any analysis population are finalized prior to unblinding. Reasons for exclusion from analysis populations are summarized by treatment group for all randomized participants and listed by participant.

#### 5.3 Analysis Populations

Analysis are based on the following study populations:

**Randomized Population:** All screened participants who provide informed consent (and assent for adolescent participants 12 to <18 years of age) and provide demographic and other screening measurements and are randomized (i.e., have a randomization number assigned within the EDC system). Most baseline summaries and the IP administration summary use the randomized population.

**Exposed Population:** All participants in the randomized population who receive IP.

**Safety Population**: All participants in the exposed population who provide safety assessment data. This generally includes any participant who was not lost to follow-up at Day 1 (baseline), as they are at risk for reporting an SAE. Participants are analyzed as treated (i.e., according to the treatment a participant received, rather than the treatment to which the participant was randomized). All safety analyses use the safety population.

**Modified Intent-to-Treat (mITT) Population**: All randomized participants who are vaccinated and have at least one post-injection anti-CHIKV human SNA assay result. Participants are counted in the group to which they were randomized. Primary and secondary

immunogenicity analyses are repeated for the mITT population as a measure of robustness of the results.

**Immunogenicity Evaluable Population (IEP):** The IEP includes all participants in the mITT population who:

- Provide evaluable serum sample results for the relevant post-vaccination time points, and within the required time frames:
  - Day 22: Day 19 through Day 27, inclusive.
- Have no measurable (≥LLOQ) anti-CHIKV human SNA assay titer at Day 1 (baseline), i.e., seronegative at baseline. Note that participants with missing Day 1 (baseline) are excluded from IEP.
- Have no important protocol deviation deemed exclusionary or other reason to be excluded as defined prior to unblinding.

The IEP is the primary population for all immunogenicity analyses.

#### 5.4 Analysis Groups

Tables are displayed by treatment group (PXVX0317 and placebo) columns with lots pooled with the exception of the lot consistency analysis, where the separate lots are displayed.

#### 5.5 Analysis Time Points

For immunogenicity analyses, anti-CHIKV SNA samples are collected at Day 1 (baseline), Day 8 (-1/+3 days), Day 15 (-1/+3 days), Day 22 (-1/+3 days) and Day 183 EOS (-14/+7 days). For the purpose of IEP membership, Day 22 has a wider window of Day 19 through Day 27, inclusive. For the time points other than the primary analysis (Day 22), all available data are included in the summaries according to the analysis set defined for a participant's inclusion.

Immunogenicity data are checked and, if another visit or unscheduled sample collection occurred closer to the nominal study day than the scheduled sample collection entered as the nominal visit, the visit data are replaced by the closer visit data when the analysis visit is assigned. In other words, the labeled database visit may not match the derived analysis visit; this procedure is necessary to mitigate the risk of data entered in an incorrect visit in the database. See also Section 5.7 describing handling of multiple sample collections in an analysis window.

Otherwise, unscheduled visit data are not presented in the by-visit summary analyses but are included in the summary tables by maximum toxicity grade or abnormality when applicable, and in data listings by participant.

#### **5.6** Definition of Baseline

For all analyses, the baseline value for each measure is defined as the last non-missing value prior to IP administration. Note that, for some participants for whom randomization system

errors delayed randomization by one calendar day, procedures performed the day before Day 1 were considered acceptable without being repeated on the actual Day 1.

#### 5.7 Multiple Records in an Analysis Window

If more than one sample is collected for anti-CHIKV human SNA assay assessment for a given time point, the sample closest to the nominal time point is used for analysis tabulations. If there is a tie (i.e., the two samples are an equidistant number of days from the nominal time point), then the geometric mean of the two titers is used for analysis tabulations. All samples are reported with database visit and analysis visit in data listings by participant.

#### **5.8** Coding Dictionaries

Medical history and AEs are coded to system organ class (SOC) and preferred term (PT) based on the Medical Dictionary for Regulatory Activities (MedDRA) dictionary version 24.1.

Prior and concomitant medications and vaccines are coded according to the World Health Organization's (WHO) WHODrug Global Dictionary version C32021 to Anatomical Therapeutic Chemical (ATC) classification and preferred drug name.

#### 5.9 Adverse Event Toxicity/Severity Grading

With the exception of redness and swelling, all solicited AEs are graded by the investigator according to severity grading scales from "mild" to "potentially life-threatening." The severity of redness and swelling, recorded as a diameter (mm) in the solicited adverse event diary, are summarized according to categories based on the largest-diameter linear measurement when a local reaction is present:

- Grade 0/absent = 0-24 mm.
- Grade 1/mild = 25-50 mm.
- Grade 2/moderate = 51-100 mm.
- Grade 3/severe = >100 mm.
- Grade 4/potentially life threatening = necrosis or exfoliative dermatitis.

Events reported as not present (0 mm is entered) are reported as Grade 0. Similarly, body temperatures recorded by the participant that are below 100.4° result in fever reported as Grade 0/absent.

Solicited AEs other than redness and swelling and unsolicited AEs are graded by the investigator for severity. The severity grading scales (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = potentially life-threatening) that are used for safety assessment in this study are provided in Appendix I of this document and Section 7.1.7 of the Protocol, based on the FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials (2). Note that AEs that result in death are classified as Grade 4 and indicated as resulting in death.

#### **6 STATISTICAL CONSIDERATIONS**

#### **6.1 Statistical Considerations**

Data summaries are tabulated by appropriate grouping for each analysis population as specified in Section 5.3.

Continuous endpoints are summarized by descriptive statistics including number of non-missing observations (n), mean, SD, median, minimum and maximum. In the analysis of the anti-CHIKV SNA data as a continuous variable, anti-CHIKV SNA values are logarithmically transformed (base10), and the GMTs and associated 95% CI for each treatment group are computed by exponentiating the corresponding log-transformed means and two-sided 95% CIs. Categorical variables are summarized by frequency counts (n) and percentages of participants (%) in each category, including missing or unknown when appropriate.

Unless otherwise specified, CIs and hypothesis tests are two-sided with 95% confidence (or one-sided with 97.5% confidence).

The reporting conventions to be applied to all tables, listings and figures are included in a living document that accompanies the table and listing shells. All derivations, statistical analyses, summaries and listings are generated using SAS Version 9.4 or higher (SAS Institute, Inc., Cary, North Carolina, United States).

#### **6.1.1** Seroresponse Rates

The superiority of the immune response to PXVX0317 vaccine over that to placebo is demonstrated at Day 22 by comparing seroresponse rates between the two treatment groups (the percentage of participants with an anti-CHIKV human SNA assay titer onsidered the presumptive seroprotection rate). Percentages of participants with anti-CHIKV SNA seroresponse rate and secondary response rates at ≥15 and 4-fold rise over baseline are reported with associated two-sided 95% Wilson score method CIs (keyword /BINOMIAL (WILSON) on tables statement). The difference in seroresponse rates between the PXVX0317 and placebo groups is calculated, along with the 95% CI for the difference based on the Newcombe hybrid score method (keyword /RISKDIFF (CL=NEWCOMBE)). The lower bound of the two-sided 95% CI on the difference in seroresponse rates between PXVX0317 and placebo must be Additionally, the null hypothesis of no difference between seroresponse rate percentages is tested using a two-sided chi-square test with alpha=0.05. No multiplicity adjustment is employed, and no covariate adjustment is performed. See Section 6.4 for statistical hypothesis, Section 6.9 for multiplicity considerations, and Section 8.4.1.1 for analysis outputs.

Identical methods will be used for treatment group comparison of seroresponse rates at Days 15, 183, and 8 as well as for lot consistency analysis of seroresponse rates.

The same methods are applied to evaluate treatment group differences in seroresponse rates at Day 22 using the composite seroresponse rate endpoint (see Section 6.3 for definition) if the baseline seropositive (anti-CHIKV SNA titer  $\geq$ LLOQ) rate is  $\geq$ 10% for the mITT population only.

#### 6.1.2 Geometric Mean Titers and Geometric Mean Fold Increase

The superiority of PXVX0317 vaccine immunogenicity over that of placebo is explored further by comparing Day 22 GMTs derived from a linear model with a one-sided alpha=0.025. The primary model is an analysis of variance (ANOVA), with log<sub>10</sub>-transformed anti-CHIKV SNA titers (log<sub>10</sub>) as the dependent variable and treatment group and study site as the fixed effects in the model. No interaction term is used. The adjusted least square means and their 95% CIs calculated based on the ANOVA are back-transformed and reported as the group GMT values. No adjustment for multiplicity is applied. See Section 6.4 for statistical hypothesis, Section 6.9 for multiplicity considerations, and Section 8.4.1.2 for analysis outputs. Identical methods are used for treatment group comparison of GMTs at Days 8, 15, and 183.

Similar methods are applied to test for a significant difference between anti-CHIKV SNA GMTs at Day 22 for PXVX0317 and placebo <u>if the baseline seropositive (SNA titer  $\geq$ LLOQ) rate is  $\geq$ 10% in the mITT population only, with baseline log-transformed SNA titer as a covariate in the ANCOVA model.</u>

GMFI from baseline (Day 1) to Days 8, 15, 22 and 183 is calculated using the difference from Day 1 in log<sub>10</sub>-transformed titers as the dependent variable in the ANOVA model. The adjusted least square means and their 95% CIs calculated based on the ANOVA are backtransformed and reported as the group GMFI values. The median, minimum and maximum titers and fold-increases are based on the non-transformed scale.

The GMTs associated with the primary lot consistency objective are also calculated via a linear model for the anti-CHIKV SNA titers collected at Day 22. The primary model is an ANOVA, with log<sub>10</sub>-transformed anti-CHIKV SNA titers as the dependent variable and vaccine lot and study site as the fixed effects in the model. No interaction term is used. The adjusted least square means and their 95% CIs calculated based on the ANOVA are backtransformed and reported as the vaccine lot GMT values. The ratio of GMTs for the comparison of the three pairs of PXVX0317 lots (A:B, B:C, A:C) is derived from this model. Pairwise equivalence testing on the log<sub>10</sub> scale uses two one-sided tests with alpha=0.025 each and no multiplicity adjustment. If for all pairs of vaccine lots, the two-sided 95% CI of the GMT ratio is within [0.667; 1.5] then lot-to-lot consistency is demonstrated. See Section 6.4 for statistical hypothesis, Section 6.9 for multiplicity considerations, and Section 8.4.1.3 for analysis outputs.

#### 6.2 Units and Precision

No intermediate rounding is performed in SDTM datasets; only final values for TFLs are rounded as follows. Immunogenicity titers are reported with one decimal place or two significant digits (e.g., 0.032, 18.0). Ratios of GMTs are presented with two decimal places.

Vital sign data are reported using standard international units. Vital signs variables including derivations thereof are reported to the same precision as the source data. Parameters derived directly from source data (e.g., minimum, maximum) or first-order statistics (e.g., mean) are reported and analyzed with the same precision as the source data. Second-order statistics (e.g., SD) are reported with one more significant digit than the source data. Percentages are reported to one decimal place.

#### **6.3** Derived Variables

This section provides definitions of the derived variables. In some cases, the definitions are provided in the relevant sections as noted.

**AE**, causing study discontinuation, is defined as a Yes response to the corresponding question on the AE eCRF.

**AE**, **medically attended (MAAE)**, is defined as a Yes response to the corresponding question on the AE eCRF.

**AE, related,** is defined as one that is "probably" or "possibly" related to IP per investigator assessment on the eCRF. If the relationship is missing for one or more occurrences of an AE for a given participant, the closest relationship of the remaining occurrences of the AE for that participant is used; if the relationship is missing for the only occurrence of an AE for a given participant, then that event is assumed to be related in order to be conservative.

**AE, resulting in death,** is defined as a Yes response to the corresponding question on the AE eCRF and/or a fatal outcome.

**AE, serious,** is defined per the derived eCRF field for AE seriousness, based on the individual criteria that make an AE qualify as serious (results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly or birth defect, or any event that may require medical or surgical intervention to prevent one of these outcomes).

**AESI** is defined in this study as new onset or worsening arthralgia that is medically attended, as noted by an AE having a Yes response to the corresponding AESI question on the AE eCRF.

**AE, severity,** is graded Grade 1 (mild) to Grade 4 (potentially life-threatening) as described in Section 5.9. If the severity is missing for one or more occurrences of an AE for a given participant, the maximum severity of the remaining occurrences of the AE for that participant is used; if the severity is missing for the only occurrence of an AE for a given participant, then that event is assumed to be severe in order to be conservative.

**AEs, solicited,** are defined as those collected in the electronic e-diary or paper diary. Solicited AEs include local (i.e., pain, redness, and swelling) and systemic reactions (i.e., fever, chills, fatigue, headache, myalgia, arthralgia, and nausea). **Solicited AEs were to be entered on Day 1 through Day 8; solicited AEs starting on Day 9 or later will be excluded from tabulations, with the exceptions of AESI and SAEs.** 

The denominator for solicited AE tables comprises only those participants with at least one diary observation (i.e., any non-missing values but excluding "Not done/unknown"), at least one diary observation for a given symptom, or at least one diary observation for a given day, as applicable. Note that an elevated in-clinic temperature assessment as part of 30-min post-vaccination vital signs does not count as a solicited AE, as vital signs data are summarized separately.

**AE**, **treatment-emergent**. AE collection begins at Day 1 (baseline), the day of IP administration. AEs occurring after a participant has given informed consent, but before vaccination, are excluded from summaries. Only treatment-emergent AEs are summarized.

AEs, unsolicited, are defined as those AEs not listed in the e-diary or paper diary but collected in the EDC. Unsolicited AEs were to be collected though Day 29 unless they were SAEs, AESI, or MAAEs; unsolicited AEs starting on Day 30 or later that are not SAEs, AESI, or MAAEs are excluded from tabulations.

**Age** at screening visit is automatically calculated by EDC based on date of birth versus date of informed consent. Age at baseline (Day 1) is be summarized in all outputs.

**Age group strata** are defined as ages 12 to <18, 18 to <46, and 46 to <65 as randomized. Note that, if a participant is randomized into a stratum and their age is later corrected such that they should have been placed into a different age stratum, the participant is analyzed according to the corrected age stratum for immunogenicity analyses.

Analysis visits are defined in Section 5.5.

Analysis populations are defined in Section 5.3.

**Baseline** is defined in Section 5.6. Change from baseline is defined as (value at post-baseline assessment – value at baseline).

**Baseline seropositive rate** is defined as the percentage of participants with anti-CHIKV human SNA assay titer ≥LLOQ.

**Body mass index** at screening visit is automatically calculated by EDC as a participant's weight in kg divided by height in m<sup>2</sup>.

Anti-chikungunya virus (anti-CHIKV) human SNA assay NT<sub>80</sub> (80% neutralizing titer) is defined as the dilution factor that corresponds to an 80% reduction of luciferase activity compared to virus-only control. Anti-CHIKV SNA titer values below LLOQ are replaced by LLOQ/2 in the immunogenicity analyses including GMT and GMFI. For the 4-fold rise over Day 1 (baseline), values below the LLOQ are replaced with the LLOQ.

**Completion of study** for an individual participant is defined as completion of the Day 183 EOS and any required safety follow-up (i.e., a disposition status of completed).

**Early discontinuation** for an individual participant is defined as completion of the Early Discontinuation/ Withdrawal Visit (i.e., a disposition status other than completed).

**Enrolled/randomized** is defined as receipt of a randomization number assignment within the EDC system.

**Lot number.** Randomization code lot letters correspond to lot numbers as follows:

- Lot 104 → A
- Lot 105 → B
- Lot  $106 \rightarrow C$

**Medical history** items entered on the medical history eCRF are considered to predate the study regardless of onset date.

**Medication, concomitant,** is defined as one taken after start of IP administration on Day 1 (baseline) through the end of study. For analysis purposes, any medication which is ongoing or with a stop date that is on or after the start date of IP administration is categorized as a concomitant medication. Partial or missing concomitant medication start and/or end date are imputed according to Section 6.5.2.

**Medication, prior,** is defined as one with a stop date within 30 days prior to the screening visit (90 days for blood products) through the start of IP administration on Day 1 (baseline).

**Protocol deviations** are defined by inclusion in the EDC protocol deviation module (participant-level only, not site-level), including monitor-identified deviations as well as Sponsor- and EDC system-identified programmatic deviations. Protocol deviations are classified by category and type (important/not important).

Randomized participant not meeting entry criteria is defined using the protocol deviation dataset and not just the inclusion exclusion criteria dataset, because a project team decision was made to keep the inclusion exclusion criteria as entered at the time of randomization even if the participant was later found to have violated entry criteria. These violations are recorded as protocol deviations.

Rounding of values is described in Section 6.2.

**Seroresponse rate** is defined as the percentage of participants who achieve an anti-CHIKV SNA titer

**Seroresponse rate, composite**, is analyzed at Day 22 if the baseline seropositive (anti-CHIKV SNA titer  $\geq$ LLOQ) rate is  $\geq$ 10%. The composite seroresponse rate endpoint is defined as follows:

- For participants seronegative at baseline (anti-CHIKV SNA titer <LLOQ), a seroresponse is defined as an anti-CHIKV SNA titer at Day 22.
- For participants seropositive at baseline (anti-CHIKV SNA titer ≥LLOQ), a seroresponse is defined as ≥4-fold rise from Day 1 (baseline) in anti-CHIKV SNA titer at Day 22.

**Study Day 1** is defined as the day of IP administration on Day 1 (baseline). The day prior to Day 1 is Day -1. There is no Day 0. If the participant is not treated, then the Day 1 (baseline) is defined as the day of randomization.

Study day relative to Day 1 are calculated as:

- Study Day = (assessment date date of Day 1 + 1) if the assessment is on or after Day 1.
- Study Day = (assessment date date of Day 1) if the assessment is before Day 1.

For conversion of durations, 1 year = 365.25 days and 1 month = 365.25/12 = 30.4375 days.

**Subgroups** for sex (male and female), race (white and non-white) and ethnicity (Hispanic or Latino and Not Hispanic or Latino) are defined based on the corresponding demographic questions. Participants missing sex, race or ethnicity will be omitted from analyses by subgroup. Participants with "Not Reported" or Unknown" ethnicity are not included in ethnicity subgroups. Product lot subgroups are defined based on the lot variable in the randomization module dataset.

Summary statistics are described in Section 6.1.

Time duration (in days) between event A and event B is (date of event B – date of event A + 1). For conversion of durations, 1 year = 365.25 days and 1 month = 365.25/12 = 30.4375 days.

**Treatment, actual,** is defined as the treatment administered to the participant by the site (i.e., corresponding to the kit number used).

**Treatment group** is defined as PXVX0317 vaccine vs. placebo.

**Treatment, randomized,** is defined as the treatment assigned to the participant by the EDC (i.e., corresponding to the kit number assigned).

#### 6.4 Statistical Hypotheses

#### 6.4.1 Coprimary Immunogenicity Endpoints

The study is a multicenter, randomized, two-arm, active-controlled study to evaluate PXVX0317 vaccine vs. placebo. A successful trial means success on each of the coprimary endpoints: seroresponse ( $H_{A1}$ ), GMT ( $H_{A2}$ ), and lot consistency pairwise GMT ratios ( $H_{A3}$ , FDA only), all at Day 22 using the IEP. Statistical hypotheses for each of these endpoints are discussed in turn in this section. The familywise error rate is fixed at a two-sided alpha of 0.05 by the requirement that all coprimary endpoints must be met for a successful outcome.

In standard statistical notation, the null and alternative hypotheses are:

H<sub>0</sub>: H<sub>A1</sub> not met or H<sub>A2</sub> not met or H<sub>A3</sub> not met

 $H_A$ :  $H_{A1}$  met and  $H_{A2}$  met and  $H_{A3}$  met

where  $H_{A1}$ ,  $H_{A2}$ , and  $H_{A3}$  are the alternative hypotheses for each of the coprimary endpoints as defined below in this section. Note:  $H_{A3}$  being met is only required for FDA.

The first coprimary endpoint is the treatment group-specific estimates and difference between treatment groups in anti-CHIKV SNA seroresponse rates using a titer of at Day 22 in the IEP for all age strata pooled and is tested in two ways. First, the lower bound of the Newcombe hybrid score method two-sided 95% CI on the difference in seroresponse rates between PXVX0317 and placebo must be secondly, the null hypothesis of no difference between seroresponse rate percentages is tested using a two-sided chi-square test with alpha=0.05. In standard statistical notation, the null and alternative hypotheses for the first coprimary endpoint are as follows:

 $H_{01}$ :  $(P_{PXVX0317} - P_{placebo})$  or  $(P_{PXVX0317} - P_{placebo}) \le 0$  using a two-sided chi-square test  $H_{A1}$ :  $(P_{PXVX0317} - P_{placebo})$  and  $(P_{PXVX0317} - P_{placebo}) > 0$  using a two-sided chi-square test where  $P_{PXVX0317}$  is the percentage of PXVX0317 participants and  $P_{placebo}$  is the percentage of placebo participants with seroresponse at a titer of  $\blacksquare$  at 21 days after vaccination in the IEP for all age strata pooled.

The second coprimary endpoint tests for a significant difference in treatment group-specific Day 22 GMTs in the IEP for all age strata pooled, as derived from a one-sided alpha=0.025

ANOVA with log<sub>10</sub>-transformed anti-CHIKV SNA titers (log<sub>10</sub>) as the dependent variable and treatment group and study site as the fixed effects. The adjusted least square means and their 95% CIs calculated based on the ANOVA are back-transformed and reported as the group GMT values. In standard statistical notation, the null and alternative hypotheses are:

```
H_{02}: (GMT_{PXVX0317} - GMT_{placebo}) \le 0
```

$$H_{A2}$$
:  $(GMT_{PXVX0317} - GMT_{placebo}) > 0$ 

where GMT<sub>PXVX0317</sub> is the GMT 21 days after vaccination for IEP participants in all age strata pooled.

The third coprimary endpoint tests the pairwise GMT ratios at Day 22 of consecutively manufactured lots (A:B, B:C, A:C) for equivalence using two one-sided tests with alpha=0.025 each in the IEP for adults 18 to <46 years of age. Pairwise GMT ratios are derived from an ANOVA model with log<sub>10</sub>-transformed anti-CHIKV SNA titers as the dependent variable and vaccine lot and study site as fixed effects. Lot-to-lot consistency is demonstrated if the two-sided 95% CI of the GMT ratio is within [0.667; 1.5] for all pairs of vaccine lots. In standard statistical notation, the null and alternative hypotheses are:

```
 \begin{array}{l} H_{03} \colon (GMT_{PXVX0317 \ lot \ A}/\ GMT_{PXVX0317 \ lot \ B}) < 0.667 \ or \\ (GMT_{PXVX0317 \ lot \ A}/\ GMT_{PXVX0317 \ lot \ B}) > 1.5 \ or \\ (GMT_{PXVX0317 \ lot \ B}/\ GMT_{PXVX0317 \ lot \ C}) < 0.667 \ or \\ (GMT_{PXVX0317 \ lot \ B}/\ GMT_{PXVX0317 \ lot \ C}) > 1.5 \ or \\ (GMT_{PXVX0317 \ lot \ A}/\ GMT_{PXVX0317 \ lot \ C}) < 0.667 \ or \\ (GMT_{PXVX0317 \ lot \ A}/\ GMT_{PXVX0317 \ lot \ C}) > 1.5 \\ H_{A3} \colon (GMT_{PXVX0317 \ lot \ A}/\ GMT_{PXVX0317 \ lot \ B}) \ge 0.667 \ and \\ (GMT_{PXVX0317 \ lot \ B}/\ GMT_{PXVX0317 \ lot \ C}) \ge 0.667 \ and \\ (GMT_{PXVX0317 \ lot \ B}/\ GMT_{PXVX0317 \ lot \ C}) \ge 0.667 \ and \\ (GMT_{PXVX0317 \ lot \ A}/\ GMT_{PXVX0317 \ lot \ C}) \ge 0.567 \ and \\ (GMT_{PXVX0317 \ lot \ A}/\ GMT_{PXVX0317 \ lot \ C}) \ge 0.567 \ and \\ (GMT_{P
```

where GMT<sub>PXVX0317 lot X</sub> is the GMT at 21 days after vaccination for IEP participants receiving PXVX0317 Lot A, B or C. Note that success on the Day 22 lot consistency endpoint is only required for FDA.

#### 6.4.2 Key Secondary Immunogenicity Endpoints

A prespecified hierarchical approach is employed for the seroresponse key secondary immunogenicity endpoints to preserve the type I error rate without the need for further multiplicity adjustment. If the null hypotheses are rejected for all coprimary endpoints, only then are the key secondary endpoints for the seroresponse rate difference (H<sub>A4</sub>) at Days 15, 183, and 8 tested sequentially, in that order, each for the IEP across all age groups combined.

At Day 15, the endpoint is tested for the success criterion of the lower bound of the two-sided Newcombe hybrid score method 95% CI on the difference in seroresponse rates between PXVX0317 and placebo and superiority to placebo is tested using a two-sided chi-square test with alpha=0.05. At Day 183 and Day 8, only superiority to placebo using a two-sided chi-square test with alpha=0.05 is tested. When a nonsignificant test is reached formal testing stops, and the remaining endpoints are reported for information only.

- 1. Day 15 seroresponse at a titer of including superiority to placebo and the success criterion of the lower bound of the two-sided Newcombe hybrid score method 95% CI on the difference in seroresponse rates between PXVX0317 and placebo
- 2. Day 183 seroresponse at a titer of including superiority to placebo.
- 3. Day 8 seroresponse at a titer of including superiority to placebo.

In standard statistical notation, the null and alternative hypotheses are:

 $H_{04}$ :  $(P_{PXVX0317} - P_{placebo})$  or  $(P_{PXVX0317} - P_{placebo}) \le 0$  using a two-sided chi-square test for Day 15 and  $(P_{PXVX0317} - P_{placebo}) \le 0$  using a two-sided chi-square test for Day 183 and Day 8.

 $H_{A4}$ :  $(P_{PXVX0317} - P_{placebo})$  and  $(P_{PXVX0317} - P_{placebo}) > 0$  using a two-sided chi-square test for Day 15 and  $(P_{PXVX0317} - P_{placebo}) > 0$  using a two-sided chi-square test for Day 183 and Day 8.

After testing the coprimary immunogenicity endpoints and, if all met, the hierarchical key secondary immunogenicity endpoints, no other formal hypothesis testing is carried out. The remaining secondary immunogenicity endpoints involving GMTs, GMFI, other titers, the exploratory endpoint, and all safety endpoints are evaluated and reported for information only, thus no further Type I error control or multiplicity adjustment is needed.

#### 6.5 Handling of Missing Data and Other Data Issues

Please see Section 6.3 for assumptions for AEs with missing relatedness and/or severity.

#### 6.5.1 Missing or Partial Dates for Solicited Adverse Events

Solicited adverse events are collected from IP administration on Day 1 until Day 8 using an electronic diary (e-diary) or backup paper diary. In the case where a participant has all eight diary entries present and a single entry is missing a date (or has a partial date), then the missing date is assumed to be the date of the missing diary entry for that participant.

# 6.5.2 Missing or Partial Dates for Unsolicited Adverse Events and Concomitant Medications

Unsolicited AE collection begins at Day 1 (baseline), the day of IP administration. *Consequently, all AEs will be considered treatment-emergent regardless of onset date.* 

For missing or partial dates for prior or concomitant medication/therapy, the following conventions are used for the purpose of determining whether the medication/therapy is concomitant or not. Original values are provided in the listings as is, without imputation.

- For start date missing completely or missing the year, impute the date to the date of first exposure to any study treatment.
- For start date missing both the month and the day, if the year is the same as the date of first exposure to any study treatment, impute the date to the date of first exposure to any study treatment, otherwise, impute the date to January 1<sup>st</sup>.
- For start date missing the day only, if the year and the month are the same as the date of first exposure to any study treatment, impute the date to the date of first exposure to any study treatment, otherwise, impute the date to the first of the month.
- For end date missing completely or missing the year, impute the date to the date of last contact.
- For end date missing both the month and the day, if the year is the same as the date of last contact, impute the date to the date of last contact, otherwise, impute the date to December 31st.
- For start date missing the day only, if the year and the month are the same as the date of last contact, impute the date to the date of last contact, otherwise, impute the date to the last day of the month.

#### **6.5.3** Missing Outcome and Covariates

Participants are included in the analyses to the extent of their available data; missing immunogenicity data are not imputed. See Sections 5.5 and 5.7 and definition of anti-CHIKV human SNA assay titer in Section 6.3.

Participants with missing categorical data are counted in missing or unknown categories when appropriate. Participants with missing numeric data are treated as missing completely at random when calculating summary statistics. For likelihood-based analyses (e.g., regression), missing at random is assumed.

#### 6.5.4 Non-Quantifiable Laboratory Data

Not applicable.

#### 6.5.5 Implausible Participant Reported Outcomes

Values measured and reported by the participant directly (e.g., via the electronic or paper diary) are not corrected in a reconciliation process. In cases where the reported values are clearly biologically implausible, the reported values and associated toxicity grades are set to missing and excluded from analysis. These reported values are included in listings.

Example: Body (oral) temperatures less than  $\leq 33^{\circ}$ C or  $\geq 42^{\circ}$ C.

#### 6.6 Adjustment for Covariates

Beyond the inclusion of site in the immunogenicity ANOVA models described in Section 6.1 and the additional inclusion of baseline log-transformed anti-CHIKV SNA titer as a covariate in the ANCOVA model if the baseline seropositive (anti-CHIKV SNA titer ≥LLOQ) rate is

 $\geq$ 10%), no further adjustment for covariates is performed. Immunogenicity analyses are conducted for all age strata pooled as well as by separate age strata.

#### 6.7 Multicenter Study

This study is expected to enroll 3150 participants at up to 50 sites in US. Data from all sites are pooled, but site is a covariate in the immunogenicity ANOVA models described in Section 6.1.

Except for lot consistency analyses, PXVX0317 lots are pooled as the PXVX0317 treatment group.

#### 6.8 Subgroup Analysis

Summaries pool all age groups and are repeated separately for each age group. Analyses of the primary immunogenicity and safety endpoints are also summarized by sex, race, and ethnicity group along with treatment group. AEs are reported by product lot subgroup.

#### 6.9 Multiplicity Adjustment

#### 6.9.1 Coprimary Immunogenicity Endpoints

The familywise error rate is fixed at a two-sided alpha of 0.05 by the requirement that all coprimary endpoints must be met for a successful outcome: seroresponse at a titer of (H<sub>A1</sub>), GMT (H<sub>A2</sub>), and lot consistency pairwise GMT ratios (H<sub>A3</sub>). See Section 6.4 for formal statistical hypotheses. Note that success on the Day 22 lot consistency endpoint is only required for FDA.

For each individual coprimary endpoint, the primary time point is Day 22 and the primary analysis population is the IEP. For the seroresponse and GMT endpoints, the primary analysis is for the pooled age strata; no multiplicity adjustment is made for the analysis of the mITT population or of the separate age strata as the primary population is the combined age groups in the IEP. For the lot consistency pairwise GMT ratios, the primary analysis is for the 18 to <46 years of age stratum; again, no multiplicity adjustment is made for the analysis of the mITT population as the primary population is the IEP.

#### 6.9.2 Key Secondary Immunogenicity Endpoints

Seroresponse key secondary immunogenicity endpoints are tested using a prespecified hierarchical strategy to preserve the type I error rate without the need for further multiplicity adjustment. These endpoints are tested formally only if the null hypotheses are rejected for all coprimary endpoints and only until a nonsignificant test is reached. If a nonsignificant test is reached formal testing stops, and the remaining endpoints are reported for information only. The sequential order of the seroresponse rate difference key secondary endpoints (H<sub>A4</sub>) is Days 15, 183, and 8, each for the IEP across all age groups combined. At Day 15, the endpoint is tested for the success criterion of the lower bound of the two-sided Newcombe hybrid score method 95% CI on the difference in seroresponse rates between PXVX0317 and

placebo and superiority to placebo using a two-sided chi-square test with alpha=0.05. At Day 183 and Day 8, only superiority to placebo using a two-sided chi-square test with alpha=0.05 is tested.

- 1. Day 15 seroresponse at a titer of including superiority to placebo and the success criterion of the lower bound of the two-sided Newcombe hybrid score method 95% CI on the difference in seroresponse rates between PXVX0317 and placebo
- 2. Day 183 seroresponse at a titer of including superiority to placebo.
- 3. Day 8 seroresponse at a titer of including superiority to placebo.

After testing the coprimary immunogenicity endpoints and, if all met, the hierarchical key secondary immunogenicity endpoints, no other formal hypothesis testing is performed. The remaining secondary immunogenicity endpoints involving GMTs, GMFI, other titers, the exploratory endpoint, and all safety endpoints are evaluated and reported for information only, thus no further multiplicity adjustment is needed.

#### 7 STUDY POPULATION CHARACTERISTICS

#### 7.1 Participant Disposition

Participant disposition over the course of the study is summarized for all randomized participants by treatment group, including number and percentages of participants still in the study each scheduled visit, competing the study and reason for not completing the study. Screen failure reasons are listed by participant. The number and percentage of participants enrolled by site are provided by treatment group for all randomized participants.

Randomization details including site, stratum, date and time of randomization, kit number, randomized treatment group assignment, and actual treatment received including lot number are listed by participant. Participants randomized but not treated, those receiving the wrong treatment, or receiving an incorrect dose are listed. Participants who were randomized despite not meeting entry criteria and those who received an excluded concomitant medication are listed

#### 7.2 Protocol Deviations

Protocol deviations defined in Section 5.1 are categorized as important or not important and evaluated for exclusion of participants from analysis populations. Important protocol deviations are tabulated by category and by treatment group for the randomized population as well as listed by participant.

#### 8 IMMUNOGENICITY ANALYSIS

#### 8.1 Populations Analyzed

The number and percentage of participants in each analysis population (randomized, exposed, safety, mITT, IEP) are summarized by treatment group for all participants. Reasons

for exclusion from analysis populations are summarized by treatment group for all randomized participants and listed by participant.

#### 8.2 Demographics and Baseline Characteristics

#### 8.2.1 Demographics

Demographic and baseline characteristics including age, age stratum, sex, race, ethnicity, baseline height, weight and body mass index, and baseline anti-CHIKV SNA serostatus (positive or negative) are tabulated by treatment group for the randomized, safety, mITT, and IEP populations for all ages pooled and by age strata. Participant site assignment is evident from the unique participant identifier.

#### **8.2.2** Baseline Disease Characteristics

This study enrolls healthy US adolescent and adult participants 12 to <65 years of age, so no baseline disease characteristics are collected.

#### 8.2.3 Medical History

Medical history is coded to the MedDRA dictionary SOC and PT (see Section 5.8). A summary table and a listing of medical history are supplied by treatment group for the randomized population.

#### 8.2.4 Prior and Concomitant Medications and Vaccines

Prior medications are defined as those taken within 30 days prior to the screening visit (90 days for blood products) through the start of IP administration on Day 1 (baseline). Concomitant medications are defined as those taken after start of IP administration on Day 1 (baseline) through the end of study. See definitions in Section 6.3. Partial dates are imputed according to Section 6.5.2.

Prior and concomitant medications and vaccines are coded to the WHODrug Global Dictionary ATC classification and preferred drug name (see Section 5.8). All prior and concomitant medications and vaccines are tabulated together by ATC classification, preferred drug name, and treatment group for the safety population; a second similar table contains only concomitant vaccines. A participant data listing of all prior and concomitant medications is generated.

#### **8.3** Treatment Compliance

As the IP administration is a single 0.8 mL intramuscular injection performed by site personnel, measurements of treatment compliance are not applicable. A vaccine administration summary is provided and details listed.

#### 8.4 Immunogenicity Analysis

Summary statistics for immunogenicity results by scheduled visit for each treatment group are provided for the IEP and mITT populations, unless otherwise specified. Anti-CHIKV SNA seroresponse rates and GMTs are tabulated by visit for each treatment group. Geometric mean fold increase as well as number and percentage of participants meeting anti-CHIKV SNA titers of ≥15 and 4-fold rise from baseline are also displayed by post-vaccination scheduled visit for each treatment group. Reverse cumulative distribution plots of anti-CHIKV SNA titer versus percentage of participants in each treatment group are generated by scheduled visit for the IEP. Anti-CHIKV SNA GMT are also plotted over time for each treatment group for the IEP.

The primary analysis of all immunogenicity endpoints utilize the IEP across all age groups combined. As specified for individual endpoints below, primary and secondary immunogenicity analyses of anti-CHIKV SNA seroresponse rates and GMTs are repeated using the mITT population as a measure of robustness of results. All immunogenicity analysis are repeated in the separate age strata for the IEP, and primary and secondary immunogenicity analyses of anti-CHIKV SNA seroresponse rates and GMTs are repeated in the separate age strata for the mITT population as well. No multiplicity adjustment is made for the analysis of the mITT population or of the separate age strata as the primary population is the combined age groups in the IEP. In addition, the primary immunogenicity endpoints using the IEP across all age groups combined are repeated by sex, by race group (white and non-white), and by ethnicity group (Hispanic or Latino and Not Hispanic or Latino).

#### 8.4.1 Coprimary Immunogenicity Endpoints

# 8.4.1.1 Day 22 Treatment Group Estimates and Difference in Anti-CHIKV SNA Seroresponse Rates

The superiority of PXVX0317 vaccine immunogenicity over that of placebo is illustrated at Day 22 by estimating the treatment-specific seroresponse rates and by calculating the difference in seroresponse rates between the two treatment groups (the percentage of participants with an anti-CHIKV SNA titer PXVX0317 minus placebo) and associated 95% CI. See Section 6.1 for statistical details.

This endpoint is summarized for all age strata pooled and for individual age strata in the IEP, as well as by sex, by race group (white and non-white), and by ethnicity group (Hispanic or Latino and Not Hispanic or Latino) for all age strata pooled in the IEP. The analysis, both for all age strata pooled and for individual age strata but not for subgroups, is repeated using the mITT population as a measure of robustness of results.

A forest plot is generated to represent seroresponse rate differences between treatment groups at Day 22 for the IEP, both for all age strata pooled and for individual age strata.

#### 8.4.1.2 Day 22 Anti-CHIKV SNA GMT by Treatment Group

Day 22 anti-CHIKV SNA GMTs and associated 95% CIs are compared between PXVX0317 and placebo treatment groups to demonstrate superiority of PXVX0317 vaccine. See Section 6.1 for statistical details.
This endpoint is summarized for all age strata pooled and for individual age strata in the IEP, as well as by sex and by race group (white and non-white) and ethnicity group (Hispanic or Latino and Not Hispanic or Latino) for all age strata pooled in the IEP. The analysis, both for all age strata pooled and for individual age strata but not for subgroups, is repeated using the mITT population as a measure of robustness of results.

A graph of anti-CHIKV SNA GMTs by visit is presented for the IEP population. As well, a reverse cumulative distribution plot of titers by visit is displayed for the IEP population.

# 8.4.1.3 Day 22 Pairwise Lot Comparison of Anti-CHIKV SNA GMT Ratio in Adults 18 to <46 years (FDA only)

The consistency of the immune response across three consecutively manufactured lots of PXVX0317 vaccine iss confirmed at Day 22 by testing equivalence of anti-CHIKV SNA GMT ratios with associated 95% CIs between all three pairs of PXVX0317 lots (A:B, A:C, B:C) among adults 18 to <46 years of age. See Section 6.1 for statistical details.

This endpoint is summarized in the IEP for the adults 18 to <46 years of age stratum only. The analysis is repeated using the mITT population for the adults 18 to <46 years of age stratum only as a measure of robustness of results.

The seroresponse rate difference (PXVX0317 minus placebo) for each vaccine lot at Day 22 is also assessed as an exploratory endpoint as described in Section 8.4.3.1.

#### 8.4.2 Secondary Immunogenicity Endpoints

# 8.4.2.1 Key Secondary Immunogenicity Endpoints: Treatment Group Estimates and Difference in Anti-CHIKV SNA Seroresponse Rates at Day 15, Day 183, and Day 8, in that order

The key secondary endpoint of treatment-specific anti-CHIKV SNA seroresponse rates and treatment group difference in seroresponse rates (PXVX0317 minus placebo) and associated 95% CI based on antibody titers measured at Day 15, Day 183, and Day 8 is analyzed as described above for Day 22. For each time point, the null hypothesis of no difference between seroresponse rate percentages in the PXVX0317 vs placebo group is tested using a chi-square test with alpha=0.05. For Day 15 only, the lower bound of the two-sided 95% CI on the difference in seroresponse rates between PXVX0317 and placebo is compared to for assessment of clinical significance.

This endpoint is summarized for all age strata pooled and for individual age strata using the IEP. The analyses are repeated using the mITT population as a measure of robustness of results.

#### 8.4.2.2 Anti-CHIKV SNA GMT at Day 8, Day 15, and Day 183 by Treatment Group

The secondary endpoint of anti-CHIKV SNA GMT and associated 95% CIs for PXVX0317 and placebo based on antibody titers measured at Day 8, Day 15, and Day 183 is analyzed as described above for Day 22.

This endpoint is summarized for all age strata pooled and for individual age strata using the IEP. The analyses are repeated using the mITT population as a measure of robustness of results.

# 8.4.2.3 GMFI in Anti-CHIKV SNA Titer from Day 1 to Days 8, 15, 22 and 183 by Treatment Group

Geometric mean fold increase over Day 1 (baseline) titer is analyzed as described for GMTs for each post-vaccination time point (Days 8, 15, 22 and 183) by treatment group. See Section 6.1 for statistical details and Section 6.3 for handling of anti-CHIKV SNA titer values below LLOQ.

This endpoint is summarized for all age strata pooled and for individual age strata using the IEP population. Geometric mean fold increase is plotted by visit for the IEP, and a reverse cumulative distribution of fold-rise from baseline by visit is also presented for the IEP.

# 8.4.2.4 Participants with Anti-CHIKV SNA Titer ≥15 and 4-fold Rise over Baseline at Days 8, 15, 22 and 183 by Treatment Group

Number and percentage of participants with an anti-CHIKV SNA titer ≥15 and 4-fold rise over Day 1 (baseline) at Days 8, 15, 22 and 183 are analyzed by treatment group as described for Day 22 seroresponse. See Section 6.1 for statistical details.

This endpoint is summarized for all age strata pooled and for individual age strata using the IEP

# 8.4.2.5 <u>If Baseline Seropositive (Anti-CHIKV SNA Titer ≥LLOQ) Rate ≥10%</u>: Treatment Group Difference in Anti-CHIKV SNA Composite Seroresponse Rate at Day 22

If the baseline seropositive (anti-CHIKV SNA titer ≥LLOQ) rate is ≥10%, difference in anti-CHIKV SNA composite seroresponse rate (PXVX0317 minus placebo) and associated 95% CI at Day 22 are analyzed for the mITT population in the same manner as described above. Composite seroresponse rate is defined in Section 6.3.

This endpoint is summarized for all age strata pooled and for individual age strata using the mITT population.

# 8.4.2.6 <u>If Baseline Seropositive (Anti-CHIKV SNA Titer ≥LLOQ) Rate ≥10%</u>: Difference in Anti-CHIKV SNA GMT at Day 22 by Treatment Group with Baseline Anti-CHIKV SNA Titer as a Covariate in the ANCOVA Model

If the baseline seropositive (anti-CHIKV SNA titer ≥LLOQ) rate is ≥10%, difference in anti-CHIKV SNA GMT and associated 95% CIs at Day 22 for PXVX0317 and placebo are analyzed using similar methods to those described above, but with baseline log-transformed anti-CHIKV SNA titer as a covariate in the ANCOVA model for the mITT population.

This endpoint is summarized for all age strata pooled and for individual age strata using the mITT population.

#### **8.4.3** Exploratory Immunogenicity Endpoints

# 8.4.3.1 Pairwise Lot Differences in Anti-CHIKV SNA Seroresponse Rate at Day 22 in Adults 18 to <46 years

Anti-CHIKV SNA seroresponse rate difference with associated 95% CIs for each pair of PXVX0317 lots (A minus B, A minus C, B minus C) is analyzed in adults 18 to <46 years of age at Day 22 in the same manner as for treatment group seroresponse rate difference. This analysis uses the IEP.

#### 8.5 Pharmacokinetic and Pharmacodynamic Analysis

Not applicable.

#### 9 SAFETY ANALYSIS

All safety data are presented in the form of tabulations and participant listings, based on the safety population.

#### 9.1 Extent of Exposure

The frequencies and percentages of participants receiving IP administration are summarized by treatment group for the randomized population, along with whether or not the dose was administered per protocol (yes/no).

#### 9.2 Adverse Events

The safety of PXVX0317 in healthy adult and adolescent participants 12 to <65 years of age is evaluated using solicited AEs occurring from IP administration on Day 1 through Day 8, unsolicited AEs through Day 29, and AESI and SAEs and MAAEs though Day 183 EOS. AEs are coded to SOC and PT according to the MedDRA dictionary per Section 5.8. They are coded for severity according to Section 5.9 and Appendix II. Only treatment-emergent AEs are summarized (i.e., excluding those after a participant has given informed consent, but before vaccination). See Section 6.3 for definitions.

Solicited AEs, unsolicited AEs, AESI and SAEs and MAAEs are summarized separately by treatment group and maximum severity for the safety population for all age strata combined. Separate participant data listings of solicited and unsolicited AEs sorted by participant identifier and AE start date are generated.

### 9.2.1 Overall Summary of Solicited and Unsolicited Adverse Events

A high-level summary of solicited and unsolicited AEs combined reviews the frequency counts and percentages of participants by treatment group reporting AEs in each of the following categories:

- Any AE and any AE ≥Grade 3
- Any solicited AE and any solicited AE ≥Grade 3

- Any treatment-related solicited AE and any treatment-related solicited AE ≥Grade 3
- Any unsolicited AE and any unsolicited AE ≥Grade 3
- Any treatment-related unsolicited AE and any treatment-related unsolicited AE ≥Grade 3
- Any SAE
- Any treatment-related SAE
- Any AE leading to study discontinuation
- Any fatal AE
- Any AESI (see definition in Section 6.3)
- Any MAAE and any treatment-related MAAE

In addition, summaries of combined solicited and unsolicited AEs by SOC, PT and highest reported severity are provided for the following populations:

- Safety population, all age groups
- Safety population by age strata
- Safety population by sex
- Safety population by race group
- Safety population by ethnicity
- Safety population by product lot

#### 9.2.2 Solicited Adverse Events from Day 1 until Day 8

Solicited AEs recorded daily in the e-diary or paper diary until Day 8 include local (i.e., pain, redness, and swelling) and systemic reactions (i.e., fever, chills, fatigue, headache, myalgia, arthralgia, and nausea). In addition, solicited AEs ongoing after seven days post-injection (Day 8) and those that are serious or MAAEs are also recorded as unsolicited AEs. Severity of solicited AEs is assessed by the investigator in the same manner as unsolicited AEs.

Frequencies and percentages of participants experiencing each solicited AE are presented by maximum severity and by treatment group. The following summaries of solicited AEs are produced:

- Solicited AEs by maximum event severity, for each event and for any event
- Solicited AEs of severe (Grade 3) or higher severity, for each event and for any event
- Treatment-related solicited AEs by maximum event severity, for each event and for any event
- Day of first onset of solicited AEs, for each event and any event
- Duration of solicited AEs, for each event and any event
- Solicited AEs by day post-injection for each event and for any event

Occurrence of at least one AE by category (local, systemic) for solicited AEs are also included.

The denominator for solicited AE tables comprises only those participants with at least one diary observation (i.e., any non-missing values but excluding "Not done/unknown"), at least one diary observation for a given symptom, or at least one diary observation for a given day, as applicable. Note that an elevated in-clinic temperature assessment as part of 30-min post-vaccination vital signs does not count as a solicited AE, as vital signs data are summarized separately.

#### 9.2.2.1 Electronic Diary Compliance

Participant compliance with e-diary or paper diary solicited adverse event entry are not summarized.

#### 9.2.3 Unsolicited Adverse Events from Day 1 through Day 29

All unsolicited AEs occurring during the specified collection period in the study are recorded, regardless of their assessment of relatedness by the investigator. Unsolicited AEs include also those solicited AEs ongoing after seven days post-injection (Day 8), AESI, and SAEs.

All reported unsolicited AEs are summarized by treatment group according to MedDRA SOC, PT and highest reported severity. When an unsolicited AE occurs more than once for a participant, the maximum severity and closest relationship to treatment is counted. The unsolicited AE analysis includes unsolicited AEs judged by the investigator as at least possibly related to IP.

#### 9.3 Deaths, Other Serious Adverse Events and Other Significant Adverse Events

#### 9.3.1 Deaths from Day 1 to Day 183 End of Study Visit

Deaths are not expected in this study with healthy participants. A tabulation and participant data listing of AEs leading to death are provided.

#### 9.3.2 Serious Adverse Events from Day 1 to Day 183 End of Study Visit

SAEs are tabulated by treatment group according to MedDRA SOC, PT and highest reported severity for all age groups and by age group stratum. A separate tabulation is limited to treatment-related SAEs only. A participant data listing of all SAEs is provided.

#### 9.3.3 Adverse Event of Special Interest from Day 1 to Day 183 End of Study Visit

AESI (see definition in Section 6.3) are tabulated by treatment group according to MedDRA SOC, PT and highest reported severity. In addition, solicited and unsolicited AESI are tabulated together.

#### 9.3.4 Medically Attended Adverse Events from Day 1 to Day 183 End of Study Visit

MAAEs (see definition in Section 6.3) are tabulated by treatment group according to MedDRA SOC, PT and highest reported severity for all age groups and by age group stratum.

## 9.3.5 Adverse Events Leading to Study Discontinuation from Day 1 to Day 183 End of Study Visit

A participant data listing of all AEs leading to study discontinuation (see definition in Section 6.3) is provided.

#### 9.3.6 Day 1 Adverse Events

A participant data listing of all AEs occurring post-vaccination on Day 1 is generated.

#### 9.4 Clinical Laboratory Tests

Not applicable.

#### 9.4.1 Pregnancy Testing

A participant listing of FSH and pregnancy test results (serum and urine) is created. A listing of pregnancy outcomes, if applicable, is provided.

#### 9.4.2 Viral Serology Testing at Screening

Viral serology testing results are supplied in a participant listing.

#### 9.5 Vital Signs, Physical Findings and Other Variables Related to Safety

#### 9.5.1 Vital Signs

Observed values in vital signs include temperature, blood pressure, respiratory rate, and heart rate at the screening visit and pre- and post-vaccination on Day 1. All vital sign records are displayed in the participant data listings.

#### 9.5.2 Physical Examinations

Physical examinations by body system include a complete examination at screening and directed examinations at Days 1, 8, 15, 22 and 183 only if indicated in order to determine if an AE needs to be recorded. Physical examination findings are listed by participant.

#### 10 DATA MONITORING AND INTERIM ANALYSIS

## 10.1 Safety Monitoring Committee

The SMC reviews aggregated, blinded safety data after the 300<sup>th</sup> enrolled participant passes Day 29, and again after the last enrolled participant passes Day 29. Refer to the separate SMC Charter for details.

### 10.2 Interim Analysis

No interim analysis is planned for this study.

#### 11 REFERENCES

- 1. CBER (2018) Guidance for Industry: Submitting Study Datasets for Vaccines to the Office of Vaccines Research and Review, Technical Specification Document.
- 2. CBER (2007) Guidance for Industry: Toxicity Grading Scale for Health Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials.
- 3. ICH E3 (1996) Guidance for Industry: Structure and Content of Clinical Study Reports.

## APPENDIX I LIST OF TABLES, FIGURES AND LISTINGS

Note the list of TFLs is a living document and subject to changes during the study.

| Table | Title |
|---|---|
| Baseline | |
| 14.1.1 | Participant Enrollment by Site – Randomized Population |
| 14.1.2 | Analysis Populations – All Participants |
| 14.1.3 | Participant Disposition – Randomized Population |
| 14.1.4.1 | Demography - Randomized Population, All Ages Pooled and by Age Group |
| 14.1.4.2 | Demography - Safety Population, All Ages Pooled and by Age Group |
| 14.1.4.3 | Demography – Modified Intent-to-treat Population, All Ages Pooled and by Age Group |
| 14.1.4.4 | Demography – Immunogenicity Evaluable Population, All Ages Pooled and by Age Group |
| 14.1.5 | Medical History – Randomized Population |
| 14.1.6 | Timing of Blood Sample Collection – Randomized Population |
| 14.1.7.1 | Important Protocol Deviations – Randomized Population |
| 14.1.7.2 | Reasons for Exclusion from Analysis Populations – Randomized Population |
| 14.1.8.1 | Prior and Concomitant Medications by Descending Frequency within ATC Class and Drug Name – Safety Population |
| 14.1.8.2 | Concomitant Vaccines by Descending Frequency within ATC Class and Drug Name – Safety Population |
| Immunogenicity | |
| 14.2.1.1.1 | Anti-CHIKV SNA Seroresponse Rate by Treatment Group and Visit – Immunogenicity Evaluable Population, All Ages Pooled and by Age Group |
| 14.2.1.1.2 | Anti-CHIKV SNA Seroresponse Rate by Treatment Group and Visit – Immunogenicity Evaluable Population, All Ages Pooled by Sex Subgroups |
| 14.2.1.1.3 | Anti-CHIKV SNA Seroresponse Rate by Treatment Group and Visit – Immunogenicity Evaluable Population, All Ages Pooled by Race Subgroups |
| 14.2.1.1.4 | Anti-CHIKV SNA Seroresponse Rate by Treatment Group and Visit – Immunogenicity Evaluable Population, All Ages Pooled by Ethnicity Subgroups |
| 14.2.1.2 | Anti-CHIKV SNA Seroresponse Rate by Treatment Group and Visit – mITT Population All Ages Pooled and by Age Group |
| 14.2.2.1.1 | Anti-CHIKV SNA GMT by Treatment Group and Visit – Immunogenicity Evaluable Population, All Ages Pooled and by Age Group |
| 14.2.2.1.2 | Anti-CHIKV SNA GMT by Treatment Group and Visit – Immunogenicity Evaluable Population, All Ages Pooled by Sex Subgroups |
| 14.2.2.1.3 | Anti-CHIKV SNA GMT by Treatment Group and Visit – Immunogenicity Evaluable Population, All Ages Pooled by Race Subgroups |
| 14.2.2.1.4 | Anti-CHIKV SNA GMT by Treatment Group and Visit – Immunogenicity Evaluable Population, All Ages Pooled by Ethnicity Subgroups |
| 14.2.2.2 | Anti-CHIKV SNA GMT by Treatment Group by Visit – mITT Population, All Ages Pooled and by Age Group |
| 14.2.3.1 | Pairwise Lot Comparison of Anti-CHIKV SNA GMT Ratio at Day 22 – Immunogenicity Evaluable Population, Adults 18 to <46 years |

| Table | Title |
|---|---|
| 14.2.3.2 | Pairwise Lot Comparison of Anti-CHIKV SNA GMT Ratio at Day 22 – mITT Population, Adults 18 to <46 years |
| 14.2.4 | Geometric Mean Fold Increase from Baseline in Anti-CHIKV SNA Titer from Day 1 to each Visit by Treatment Group – Immunogenicity Evaluable Population, All Ages Pooled and by Age Group |
| 14.2.5 | Participants with Anti-CHIKV SNA at or above Selected Titers by Treatment Group and Visit – Immunogenicity Evaluable Population, All Ages Pooled and by Age Group |
| 14.2.6 | Pairwise Lot Comparison of Anti-CHIKV SNA Seroresponse Rate at Day 22 – Immunogenicity Evaluable Population, Adults 18 to <46 years |
| 14.2.7 | If Baseline Seropositive Rate ≥10%: Anti-CHIKV SNA Composite Seroresponse Rate at Day 22 by Treatment Group – mITT Population, All Ages Pooled and by Age Group |
| 14.2.8 | If Baseline Seropositive Rate ≥10%: Anti-CHIKV SNA GMT at Day 22 by Treatment Group with Baseline Titer as a Covariate – mITT Population, All Ages Pooled and by Age Group |
| Safety | |
| 14.3.1 | Vaccine Administration – Randomized Population |
| 14.3.2.1 | High Level Summary of Solicited and Unsolicited Adverse Events – Safety Population, All Ages Pooled |
| 14.3.2.2.1 | Solicited Adverse Events by Highest Reported Severity – Safety Population, All Ages Pooled and by Age Group |
| 14.3.2.2.2 | Solicited Adverse Events by Highest Reported Severity – Safety Population, All Ages Pooled by Sex Subgroups |
| 14.3.2.2.3 | Solicited Adverse Events by Highest Reported Severity – Safety Population, All Ages Pooled by Race Subgroups |
| 14.3.2.2.4 | Solicited Adverse Events by Highest Reported Severity – Safety Population, All Ages Pooled by Ethnicity Subgroups |
| 14.3.2.3 | Solicited Events of Severe (Grade 3) or Higher Severity by Highest Reported Severity – Safety Population, All Ages Pooled |
| 14.3.2.4 | Treatment-related Solicited Adverse Events by Highest Reported Severity – Safety Population, All Ages Pooled |
| 14.3.2.5.1 | Day of Onset for Participants who Reported Solicited Adverse Events – Safety Population, All Ages Pooled |
| 14.3.2.5.2 | Day of Onset for Participants who Reported Treatment-related Solicited Adverse Events – Safety Population, All Ages Pooled |
| 14.3.2.6.1 | Number of Days with Symptoms for Participants who Reported Solicited Adverse Events – Safety Population, All Ages Pooled |
| 14.3.2.6.2 | Number of Days with Symptoms for Participants who Reported Treatment-related Solicited Adverse Events – Safety Population, All Ages Pooled |
| 14.3.2.7 | Percentage of Participants with Solicited Adverse Events by Day on Study – Safety Population, All Ages Pooled |
| 14.3.3.1 | Solicited and Unsolicited Adverse Events by System Organ Class, Preferred Term and Highest Reported Severity – Safety Population, All Ages Pooled and by Age Group |
| 14.3.3.2 | Solicited and Unsolicited Adverse Events by Highest Reported Severity – Safety Population by Sex Subgroups |
| 14.3.3.3 | Solicited and Unsolicited Adverse Events by Highest Reported Severity – Safety Population by Race Subgroups |

| Table | Title |
|---|---|
| 14.3.3.4 | Solicited and Unsolicited Adverse Events by Highest Reported Severity – Safety Population by Ethnicity Subgroups |
| 14.3.3.5 | Solicited and Unsolicited Adverse Events Excluding Serious Adverse Events by System Organ Class, Preferred Term and Highest Reported Severity – Safety Population, All Ages Pooled |
| 14.3.4.1 | Listing of Serious Adverse Events - Safety Population, All Ages Pooled |
| 14.3.4.2 | Listing of Adverse Events Leading to Study Discontinuation – Safety Population, All Ages Pooled |
| 14.3.4.3 | Listing of Adverse Events Leading to Death - Safety Population, All Ages Pooled |
| 14.3.5.1 | Unsolicited Adverse Events in Descending Frequency by Preferred Term – Safety Population, All Ages Pooled |
| 14.3.5.2 | Unsolicited Adverse Events by System Organ Class, Preferred Term and Highest Reported Severity – Safety Population, All Ages Pooled and by Age Group |
| 14.3.5.3 | Unsolicited Adverse Events of Severe (Grade 3) or Higher Severity in Descending Frequency by Preferred Term – Safety Population, All Ages Pooled |
| 14.3.5.4 | Unsolicited Adverse Events of Severe (Grade 3) or Higher Severity by System Organ Class, Preferred Term and Highest Reported Severity – Safety Population, All Ages Pooled |
| 14.3.5.5 | Treatment-related Unsolicited Adverse Events in Descending Frequency by Preferred Term – Safety Population, All Ages Pooled |
| 14.3.5.6 | Treatment-related Unsolicited Adverse Events by System Organ Class, Preferred Term and Highest Reported Severity – Safety Population, All Ages Pooled |
| 14.3.5.7 | Serious Adverse Events by System Organ Class, Preferred Term and Highest Reported Severity – Safety Population, All Ages Pooled and by Age Group |
| 14.3.5.8 | Treatment-related Serious Adverse Events by System Organ Class, Preferred Term and Highest Reported Severity – Safety Population, All Ages Pooled |
| 14.3.5.9 | Adverse Events of Special Interest by System Organ Class, Preferred Term and Highest Reported Severity – Safety Population, All Ages Pooled |
| 14.3.5.10 | Adverse Events of Special Interest Including Solicited Events by System Organ Class, Preferred Term and Highest Reported Severity – Safety Population, All Ages Pooled |
| 14.3.5.11 | Medically Attended Adverse Events by System Organ Class, Preferred Term and Highest Reported Severity – Safety Population, All Ages Pooled and by Age Group |
| 14.3.5.12 | Treatment-related Medically Attended Adverse Events by System Organ Class, Preferred Term and Highest Reported Severity – Safety Population, All Ages Pooled |

| Figure | Title |
|---|---|
| 14.4.2.1.1 | Forest Plot of Seroresponse Rate at Day 22 – Immunogenicity Evaluable Population, All Ages Pooled and by Age Group |
| 14.4.2.1.2 | Forest Plot of Seroresponse Rate at Day 22 – Immunogenicity Evaluable Population, All Ages Pooled by Sex, Race, and Ethnicity Subgroups |
| 14.4.2.2.1 | Geometric Mean Anti-CHIKV SNA Titers by Visit – Immunogenicity Evaluable Population, All Ages Pooled |
| 14.4.2.2.2 | Reverse Cumulative Distribution of Anti-CHIKV SNA Titers by Visit – Immunogenicity Evaluable Population, All Ages Pooled |

| Figure | Title |
|---|---|
| 14.4.2.1.1 | Forest Plot of Seroresponse Rate at Day 22 – Immunogenicity Evaluable Population, All Ages Pooled and by Age Group |
| 14.4.2.1.2 | Forest Plot of Seroresponse Rate at Day 22 – Immunogenicity Evaluable Population, All Ages Pooled by Sex, Race, and Ethnicity Subgroups |
| 14.4.2.2.1 | Geometric Mean Anti-CHIKV SNA Titers by Visit – Immunogenicity Evaluable Population, All Ages Pooled |
| 14.4.2.3.1 | Geometric Mean Fold Increase in Anti-CHIKV SNA Titers by Visit – Immunogenicity Evaluable Population, All Ages Pooled |
| 14.4.2.3.2 | Reverse Cumulative Distribution of Geometric Mean Fold Increase in Anti-CHIKV SNA Titers by Visit – Immunogenicity Evaluable Population, All Ages Pooled |

| Listing | Title |
|---|---|
| 16.1.6 and | |
| 16.1.7 | Participant Randomization Assignments |
| 16.2.1.1 | Participant Disposition |
| 16.2.1.2 | Reasons for Screen Failure |
| 16.2.2.1 | Participants Randomized who Did Not Satisfy Entry Criteria |
| 16.2.2.2 | Participants who Received the Wrong Treatment or an Incorrect Dose |
| 16.2.2.3 | Participants who Received an Excluded Concomitant Medication |
| 16.2.2.4 | Important Protocol Deviations |
| 16.2.3 | Analysis Populations |
| 16.2.4.1 | Demography |
| 16.2.4.2.1 | Medical History |
| 16.2.4.2.2 | Verbatim to Preferred Term Mapping for Medical History |
| 16.2.4.3 | Prior and Concomitant Medications and Vaccines |
| 16.2.4.4 | Verbatim to Preferred Name Mapping for Concomitant Medications |
| 16.2.5 | Anti-CHIKV SNA Titers |
| 16.2.6 | Study Vaccine Administration |
| 16.2.7.1 | Solicited Adverse Events |
| 16.2.7.2.1 | Unsolicited Adverse Events |
| 16.2.7.2.2 | Unsolicited Adverse Events Occurring Postvaccination on Day 1 |
| 16.2.7.3 | Verbatim to Preferred Term Mapping for Unsolicited Adverse Events |
| 16.2.7.4 | Participant Identification of Adverse Events |
| 16.2.8.1 | Vital Sign Results |
| 16.2.8.2 | Physical Examination Results |
| 16.2.8.3.1 | Pregnancy Test Results |
| 16.2.8.3.2 | Pregnancy Outcomes |
| 16.2.8.4 | Viral Screening Results |
| 16.2.8.5 | Hospitalization Details |
| 16.2.8.6 | Death Details |

### APPENDIX II TOXICITY GRADING SCALE

| EVENT | MILD<br>(Grade 1) | MODERATE<br>(Grade 2) | SEVERE<br>(Grade 3) | POTENTIALLY<br>LIFE<br>THREATENING<br>(Grade 4) |
|---|---|---|---|---|
| Fever | ≥100.4-101.1°F<br>(≥38.0-38.4°C) | ≥101.2-102°F<br>(≥38.5-<39°C) | ≥102.1°F-104°F<br>(≥39°C-40°C) | >104°F<br>(>40°C) |
| Headache | No interference with activity | Some interference with activity, may require repeated use of non-narcotic pain reliever for more than 24 hours | Significant,<br>prevents daily<br>activity, any use<br>of narcotic pain<br>reliever | ER visit or<br>hospitalization |
| Fatigue | No interference with activity | Some interference with activity | Significant, prevents daily activity | ER visit or hospitalization |
| Myalgia | No interference with activity | Some interference with activity | Significant, prevents daily activity | ER visit or hospitalization |
| Nausea | No interference with activity | Some interference with activity | Significant, prevents daily activity | ER visit or<br>hospitalization for<br>hypotensive shock |
| Vomiting | 1–2 episodes/24 hours | >2 episodes/24<br>hours | Requires IV hydration | ER visit or<br>hospitalization for<br>hypotensive shock |
| Diarrhea | 2-3 loose stools<br>or <400 g/24<br>hours | 4-5 stools or 400-<br>800 g/24 hours | 6 or more<br>watery stools or<br>>800 g/24 hours<br>or requires<br>outpatient IV<br>hydration | ER visit or<br>hospitalization |
| Injection site pain | Does not interfere with activity | Repeated use of<br>non-narcotic pain<br>reliever > 24 hours<br>or interferes with<br>activity | Use of any<br>narcotic pain<br>reliever or<br>prevents daily<br>activity | ER visit or hospitalization |
| Injection site erythema/redness | 25-50 mm | 51 mm-100 mm | >100 mm | Necrosis or exfoliative dermatitis |
| Injection site induration/swelling | 25-50 mm<br>and does not<br>interfere with<br>activity | 51 mm-100 mm<br>or interferes with<br>activity | >100 mm<br>or prevents daily<br>activity | Necrosis |

## Document Approvals Approved Date: 27 Mar 2023

| Document Approval Task<br>Verdict: Approve | Director, Biostatistics |
|---|---|
| Document Approval Task<br>Verdict: Approve | Sr Director, Biostatistics & Data Sciences |
| Document Approval Task<br>Verdict: Approve | Sr. Manager, Clinical Trials |
| Document Approval Task<br>Verdict: Approve | VP, Clinical Development |